CLINICAL TRIAL: NCT03563183
Title: Observational Study to Assess Frailty of Subjects During ZOSTER-006 and ZOSTER-022 and HZ Efficacy, Immunogenicity and Safety of HZ/su by Frailty Status
Brief Title: A Study to Assess Frailty of Subjects During ZOSTER-006 and ZOSTER-022
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 204878
Record Dates: First submitted 2018-06-04; First posted 2018-06-20 (Actual); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Herpes Zoster
Keywords: immunogenicity; Herpes Zoster; efficacy; safety; frailty; Shingles vaccine
MeSH Terms: conditions — Herpes Zoster; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Overall Group: Adults aged ≥50 years of age in the Zoster-064 TVC who received herpes zoster subunit (HZ/su) vaccine or Placebo in Zoster-006/022 study
  Interventions: Other: Encoding of data collected in Zoster 006 and Zoster 022 studies

INTERVENTIONS:
Other: Encoding of data collected in Zoster 006 and Zoster 022 studies — Not applicable (disease epidemiology study)

SUMMARY:
As part of the ZOSTER-006 and ZOSTER-022 pivotal trials of the HZ/su vaccine, all study participants completed quality of life (QoL) questionnaires. The only questionnaires encoded into the data base were those from participants who developed a suspected shingles episode during the study.

The purpose of this study is to allow for the encoding and analysis of questionnaires for all subjects enrolled in ZOSTER-006 and ZOSTER-022. The aim is to assess the baseline frailty of subjects enrolled in these studies and to investigate whether this population is representative of the general population.

DETAILED DESCRIPTION:
As part of the study procedure, each subject enrolled in studies Zoster-006 and Zoster-022 was asked to complete two quality of life (QoL) questionnaires named respectively SF-36 and EQ-5D at predefined study time points. These questionnaires were to provide relevant information about the quality of life (functional status, ability to socialize, mental health, etc.) of subjects before they develop shingles Extracting some elements of the Quality of Life questionnaires (QoL), EQ-5D and SF-36, completed by all study subjects at baseline, and combining them with other medical history data allows attributing of frailty scores.

Analyses pertaining to efficacy, safety and immunogenicity as per frailty score might be performed according to the methodology used in the ZOSTER-006 and ZOSTER-022 studies.

Additionally, the data collected can be used to assess if some physical, physiological and/or psychological characteristics reported by the subjects before the onset of HZ would be predictive of HZ.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who participated in the Zoster 006 and Zoster 022 trials.
* Subjects who died or were lost to follow-up during ZOSTER-006 and ZOSTER-022 will be considered for enrolment in ZOSTER-064 and their data/questionnaires up to that point will be used.

Exclusion Criteria:

* Subjects who were excluded from all analyses from ZOSTER-006 and ZOSTER-022. This will include any subject eliminated following deviations from GCP compliance.
* Subjects who developed a suspected HZ case during ZOSTER-006 and ZOSTER-022 (since their QoL questionnaires were encoded in the eCRF for ZOSTER-006 and ZOSTER-022).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects enrolled in the Zoster 006 and Zoster 022 studies
Sampling Method: Non-Probability Sample
Enrollment: 26976 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (144):
- United States (29):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Mt Pleasant, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Beachwood, Ohio
  - GSK Investigational Site, Wadsworth, Ohio
  - GSK Investigational Site, Pleasant Hills, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Winchester, Virginia
  - GSK Investigational Site, Renton, Washington
- Australia (5):
  - GSK Investigational Site, Maroubra, New South Wales
  - GSK Investigational Site, Umina, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Sherwood, Queensland
- Brazil (4):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Curitiba/PR
  - GSK Investigational Site, São Paulo
- Canada (12):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Woodstock, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- GSK Investigational Site, Hradec Králové, Czechia
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- GSK Investigational Site, Tampereen Yliopisto, Finland
- France (13):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Château-Gontier
  - GSK Investigational Site, Cherbourg
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Montrevault
  - GSK Investigational Site, Muret
  - GSK Investigational Site, Mûrs-Erigné
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Rosiers-d'Égletons
  - GSK Investigational Site, Saint-Cyr-sur-Loire
  - GSK Investigational Site, Segré
  - GSK Investigational Site, Tours
- Germany (29):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Dachau, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Rednitzhembach, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Flörsheim, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Duelmen, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Magdeburg
- Hong Kong (2):
  - GSK Investigational Site, Kwun Tong
  - GSK Investigational Site, Shatin
- Italy (6):
  - GSK Investigational Site, Chieti, Abruzzo
  - GSK Investigational Site, Pescara, Abruzzo
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Monza, Lombardy
  - GSK Investigational Site, Cuneo, Piedmont
- Japan (3):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Tokyo
- Mexico (2):
  - GSK Investigational Site, Zapopan, Jalisco, Jalisco
  - GSK Investigational Site, Durango
- South Korea (4):
  - GSK Investigational Site, Gangwon-do
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (11):
  - GSK Investigational Site, Alcover( Tarragona)
  - GSK Investigational Site, Balenyà (Barcelona)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda( Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Peralada( Girona)
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vic/ Barcelona
- Sweden (10):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Uppsala
  - GSK Investigational Site, Vällingby
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan
- United Kingdom (7):
  - GSK Investigational Site, Atherstone, Warwickshire
  - GSK Investigational Site, Bradford-on-Avon, Wiltshire
  - GSK Investigational Site, Bangor
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Broughshane
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Newtonabbey

REFERENCES:
- [Derived] Curran D, Kim JH, Matthews S, Dessart C, Levin MJ, Oostvogels L, Riley ME, Schmader KE, Cunningham AL, McNeil SA, Schuind AE, Andrew MK; Zoster-064 Study Group. Recombinant Zoster Vaccine Is Efficacious and Safe in Frail Individuals. J Am Geriatr Soc. 2021 Mar;69(3):744-752. doi: 10.1111/jgs.16917. Epub 2020 Nov 16. PMID 33197294

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 29305 subjects in the Total Vaccinated cohort (TVC) of study ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229), 2329 subjects were excluded as they belonged to centers not participating in the current study Zoster-064(Z-064). Thus, 26976 subjects were eligible for Inclusion in the Z-064 TVC.
Period: Overall Study
Arm/Group | Overall Group
Started | 26976
Completed | 26976
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Group
Number analyzed (Participants) | 26976
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15685
  Male | 11291
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 347
  American Indian or Alaskan Native | 20
  Asian - Central/South Asian Heritage | 13
  Asian - East Asian Heritage | 4090
  Asian - Japanese Heritage | 901
  Asian - South East Asian Heritage | 38
  Native Hawaiian or Other Pacific Islander | 6
  White - Arabic / North African Heritage | 161
  White - Caucasian / European Heritage | 20112
  Other | 1288

OUTCOME MEASURES:

1. Secondary Outcome: Distribution of Short Form 36 (SF-36) Questionnaire Scale Scores, by Country
Description: The mean and standard deviation of the SF-36 Questionnaire scale scores are presented for each time point. The SF-36 is a multi-purpose health survey with 36 questions underlying the construction of 8 scales [Ware, 2001]: Physical Functioning (PF), Role Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Emotional (RE) and Mental Health (MH).
  All but one of the 36 items (self-reported health transition) are used to score the eight SF-36 scales. Each item is used in scoring only one scale. Scale scores are constructed following the summated ratings and standardized SF-36 scoring algorithms. The SF-36 scores range from 0 to 100, with high scores indicating high levels of functioning/quality of life.
Time Frame: At Month 0, 14, 26 and 38
Population: Analysis was performed on all subjects included in the Total Vaccinated Cohort (TVC) of Zoster-064
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Overall Group
Number analyzed (Participants) | 26976
Scale score
  Month 0 - SF36 PF (Australia): number analyzed (Participants) | 481
  Month 0 - SF36 PF (Australia) | 75.50 (23.366)
  Month 0 - SF36 RP (Australia): number analyzed (Participants) | 481
  Month 0 - SF36 RP (Australia) | 80.43 (24.521)
  Month 0 - SF36 BP (Australia): number analyzed (Participants) | 481
  Month 0 - SF36 BP (Australia) | 74.49 (23.545)
  Month 0 - SF36 GH (Australia): number analyzed (Participants) | 481
  Month 0 - SF36 GH (Australia) | 76.15 (17.016)
  Month 0 - SF36 VT (Australia): number analyzed (Participants) | 481
  Month 0 - SF36 VT (Australia) | 67.58 (18.344)
  Month 0 - SF36 SF (Australia): number analyzed (Participants) | 481
  Month 0 - SF36 SF (Australia) | 91.11 (16.485)
  Month 0 - SF36 RE (Australia): number analyzed (Participants) | 481
  Month 0 - SF36 RE (Australia) | 88.76 (19.879)
  Month 0 - SF36 MH (Australia): number analyzed (Participants) | 481
  Month 0 - SF36 MH (Australia) | 84.12 (13.975)
  Month 14 - SF36 PF (Australia): number analyzed (Participants) | 436
  Month 14 - SF36 PF (Australia) | 72.78 (24.472)
  Month 14 - SF36 RP (Australia): number analyzed (Participants) | 436
  Month 14 - SF36 RP (Australia) | 76.39 (26.339)
  Month 14 - SF36 BP (Australia): number analyzed (Participants) | 435
  Month 14 - SF36 BP (Australia) | 70.46 (24.483)
  Month 14 - SF36 GH (Australia): number analyzed (Participants) | 437
  Month 14 - SF36 GH (Australia) | 71.73 (18.227)
  Month 14 - SF36 VT (Australia): number analyzed (Participants) | 435
  Month 14 - SF36 VT (Australia) | 64.26 (21.926)
  Month 14 - SF36 SF (Australia): number analyzed (Participants) | 436
  Month 14 - SF36 SF (Australia) | 85.92 (23.581)
  Month 14 - SF36 RE (Australia): number analyzed (Participants) | 436
  Month 14 - SF36 RE (Australia) | 86.07 (22.532)
  Month 14 - SF36 MH (Australia): number analyzed (Participants) | 435
  Month 14 - SF36 MH (Australia) | 82.18 (16.909)
  Month 26 - SF36 PF (Australia): number analyzed (Participants) | 412
  Month 26 - SF36 PF (Australia) | 73.01 (24.468)
  Month 26 - SF36 RP (Australia): number analyzed (Participants) | 412
  Month 26 - SF36 RP (Australia) | 76.12 (25.386)
  Month 26 - SF36 BP (Australia): number analyzed (Participants) | 412
  Month 26 - SF36 BP (Australia) | 70.10 (24.188)
  Month 26 - SF36 GH (Australia): number analyzed (Participants) | 413
  Month 26 - SF36 GH (Australia) | 70.38 (18.815)
  Month 26 - SF36 VT (Australia): number analyzed (Participants) | 412
  Month 26 - SF36 VT (Australia) | 62.18 (21.385)
  Month 26 - SF36 SF (Australia): number analyzed (Participants) | 412
  Month 26 - SF36 SF (Australia) | 87.26 (21.499)
  Month 26 - SF36 RE (Australia): number analyzed (Participants) | 412
  Month 26 - SF36 RE (Australia) | 85.84 (22.472)
  Month 26 - SF36 MH (Australia): number analyzed (Participants) | 412
  Month 26 - SF36 MH (Australia) | 81.22 (17.017)
  Month 38 - SF36 PF (Australia): number analyzed (Participants) | 403
  Month 38 - SF36 PF (Australia) | 71.83 (25.972)
  Month 38 - SF36 RP (Australia): number analyzed (Participants) | 403
  Month 38 - SF36 RP (Australia) | 74.16 (27.235)
  Month 38 - SF36 BP (Australia): number analyzed (Participants) | 403
  Month 38 - SF36 BP (Australia) | 70.06 (23.919)
  Month 38 - SF36 GH (Australia): number analyzed (Participants) | 403
  Month 38 - SF36 GH (Australia) | 70.79 (19.777)
  Month 38 - SF36 VT (Australia): number analyzed (Participants) | 402
  Month 38 - SF36 VT (Australia) | 63.68 (21.220)
  Month 38 - SF36 SF (Australia): number analyzed (Participants) | 403
  Month 38 - SF36 SF (Australia) | 86.14 (21.822)
  Month 38 - SF36 RE (Australia): number analyzed (Participants) | 403
  Month 38 - SF36 RE (Australia) | 85.57 (22.371)
  Month 38 - SF36 MH (Australia): number analyzed (Participants) | 402
  Month 38 - SF36 MH (Australia) | 82.26 (15.807)
  Month 0 - SF36 PF (Brazil): number analyzed (Participants) | 1252
  Month 0 - SF36 PF (Brazil) | 74.90 (23.505)
  Month 0 - SF36 RP (Brazil): number analyzed (Participants) | 1255
  Month 0 - SF36 RP (Brazil) | 81.74 (24.185)
  Month 0 - SF36 BP (Brazil): number analyzed (Participants) | 1253
  Month 0 - SF36 BP (Brazil) | 69.57 (26.057)
  Month 0 - SF36 GH (Brazil): number analyzed (Participants) | 1255
  Month 0 - SF36 GH (Brazil) | 76.25 (18.983)
  Month 0 - SF36 VT (Brazil): number analyzed (Participants) | 1250
  Month 0 - SF36 VT (Brazil) | 72.53 (20.835)
  Month 0 - SF36 SF (Brazil): number analyzed (Participants) | 1255
  Month 0 - SF36 SF (Brazil) | 84.33 (21.505)
  Month 0 - SF36 RE (Brazil): number analyzed (Participants) | 1250
  Month 0 - SF36 RE (Brazil) | 83.48 (22.963)
  Month 0 - SF36 MH (Brazil): number analyzed (Participants) | 1251
  Month 0 - SF36 MH (Brazil) | 79.13 (19.192)
  Month 14 - SF36 PF (Brazil): number analyzed (Participants) | 1149
  Month 14 - SF36 PF (Brazil) | 72.60 (23.984)
  Month 14 - SF36 RP (Brazil): number analyzed (Participants) | 1148
  Month 14 - SF36 RP (Brazil) | 79.01 (26.311)
  Month 14 - SF36 BP (Brazil): number analyzed (Participants) | 1150
  Month 14 - SF36 BP (Brazil) | 68.14 (26.068)
  Month 14 - SF36 GH (Brazil): number analyzed (Participants) | 1151
  Month 14 - SF36 GH (Brazil) | 74.10 (19.110)
  Month 14 - SF36 VT (Brazil): number analyzed (Participants) | 1150
  Month 14 - SF36 VT (Brazil) | 71.70 (21.709)
  Month 14 - SF36 SF (Brazil): number analyzed (Participants) | 1150
  Month 14 - SF36 SF (Brazil) | 83.22 (23.396)
  Month 14 - SF36 RE (Brazil): number analyzed (Participants) | 1150
  Month 14 - SF36 RE (Brazil) | 84.07 (23.233)
  Month 14 - SF36 MH (Brazil): number analyzed (Participants) | 1150
  Month 14 - SF36 MH (Brazil) | 78.24 (20.318)
  Month 26 - SF36 PF (Brazil): number analyzed (Participants) | 1118
  Month 26 - SF36 PF (Brazil) | 73.28 (24.185)
  Month 26 - SF36 RP (Brazil): number analyzed (Participants) | 1117
  Month 26 - SF36 RP (Brazil) | 81.85 (25.360)
  Month 26 - SF36 BP (Brazil): number analyzed (Participants) | 1116
  Month 26 - SF36 BP (Brazil) | 69.69 (26.737)
  Month 26 - SF36 GH (Brazil): number analyzed (Participants) | 1118
  Month 26 - SF36 GH (Brazil) | 74.96 (19.553)
  Month 26 - SF36 VT (Brazil): number analyzed (Participants) | 1117
  Month 26 - SF36 VT (Brazil) | 71.92 (21.804)
  Month 26 - SF36 SF (Brazil): number analyzed (Participants) | 1117
  Month 26 - SF36 SF (Brazil) | 85.78 (22.726)
  Month 26 - SF36 RE (Brazil): number analyzed (Participants) | 1116
  Month 26 - SF36 RE (Brazil) | 85.78 (21.389)
  Month 26 - SF36 MH (Brazil): number analyzed (Participants) | 1117
  Month 26 - SF36 MH (Brazil) | 79.57 (19.974)
  Month 38 - SF36 PF (Brazil): number analyzed (Participants) | 1094
  Month 38 - SF36 PF (Brazil) | 71.21 (25.322)
  Month 38 - SF36 RP (Brazil): number analyzed (Participants) | 1095
  Month 38 - SF36 RP (Brazil) | 80.08 (26.268)
  Month 38 - SF36 BP (Brazil): number analyzed (Participants) | 1095
  Month 38 - SF36 BP (Brazil) | 68.77 (26.803)
  Month 38 - SF36 GH (Brazil): number analyzed (Participants) | 1095
  Month 38 - SF36 GH (Brazil) | 73.18 (20.140)
  Month 38 - SF36 VT (Brazil): number analyzed (Participants) | 1095
  Month 38 - SF36 VT (Brazil) | 70.61 (20.626)
  Month 38 - SF36 SF (Brazil): number analyzed (Participants) | 1095
  Month 38 - SF36 SF (Brazil) | 83.81 (22.055)
  Month 38 - SF36 RE (Brazil): number analyzed (Participants) | 1095
  Month 38 - SF36 RE (Brazil) | 84.27 (22.853)
  Month 38 - SF36 MH (Brazil): number analyzed (Participants) | 1095
  Month 38 - SF36 MH (Brazil) | 77.96 (20.046)
  Month 0 - SF36 PF (Canada): number analyzed (Participants) | 1365
  Month 0 - SF36 PF (Canada) | 76.09 (23.037)
  Month 0 - SF36 RP (Canada): number analyzed (Participants) | 1385
  Month 0 - SF36 RP (Canada) | 80.66 (23.449)
  Month 0 - SF36 BP (Canada): number analyzed (Participants) | 1365
  Month 0 - SF36 BP (Canada) | 75.10 (23.078)
  Month 0 - SF36 GH (Canada): number analyzed (Participants) | 1386
  Month 0 - SF36 GH (Canada) | 78.52 (16.334)
  Month 0 - SF36 VT (Canada): number analyzed (Participants) | 1384
  Month 0 - SF36 VT (Canada) | 71.69 (16.811)
  Month 0 - SF36 SF (Canada): number analyzed (Participants) | 1385
  Month 0 - SF36 SF (Canada) | 91.16 (16.701)
  Month 0 - SF36 RE (Canada): number analyzed (Participants) | 1384
  Month 0 - SF36 RE (Canada) | 88.48 (19.363)
  Month 0 - SF36 MH (Canada): number analyzed (Participants) | 1384
  Month 0 - SF36 MH (Canada) | 83.37 (14.410)
  Month 14 - SF36 PF (Canada): number analyzed (Participants) | 1341
  Month 14 - SF36 PF (Canada) | 73.53 (25.628)
  Month 14 - SF36 RP (Canada): number analyzed (Participants) | 1341
  Month 14 - SF36 RP (Canada) | 77.13 (25.882)
  Month 14 - SF36 BP (Canada): number analyzed (Participants) | 1339
  Month 14 - SF36 BP (Canada) | 72.65 (24.338)
  Month 14 - SF36 GH (Canada): number analyzed (Participants) | 1341
  Month 14 - SF36 GH (Canada) | 75.14 (18.174)
  Month 14 - SF36 VT (Canada): number analyzed (Participants) | 1338
  Month 14 - SF36 VT (Canada) | 68.40 (19.040)
  Month 14 - SF36 SF (Canada): number analyzed (Participants) | 1339
  Month 14 - SF36 SF (Canada) | 87.72 (19.983)
  Month 14 - SF36 RE (Canada): number analyzed (Participants) | 1341
  Month 14 - SF36 RE (Canada) | 85.55 (22.416)
  Month 14 - SF36 MH (Canada): number analyzed (Participants) | 1338
  Month 14 - SF36 MH (Canada) | 81.57 (15.655)
  Month 26 - SF36 PF (Canada): number analyzed (Participants) | 1286
  Month 26 - SF36 PF (Canada) | 72.97 (25.430)
  Month 26 - SF36 RP (Canada): number analyzed (Participants) | 1292
  Month 26 - SF36 RP (Canada) | 76.35 (25.745)
  Month 26 - SF36 BP (Canada): number analyzed (Participants) | 1286
  Month 26 - SF36 BP (Canada) | 71.62 (23.950)
  Month 26 - SF36 GH (Canada): number analyzed (Participants) | 1292
  Month 26 - SF36 GH (Canada) | 74.86 (18.540)
  Month 26 - SF36 VT (Canada): number analyzed (Participants) | 1292
  Month 26 - SF36 VT (Canada) | 67.67 (19.021)
  Month 26 - SF36 SF (Canada): number analyzed (Participants) | 1292
  Month 26 - SF36 SF (Canada) | 87.83 (19.836)
  Month 26 - SF36 RE (Canada): number analyzed (Participants) | 1290
  Month 26 - SF36 RE (Canada) | 85.08 (22.514)
  Month 26 - SF36 MH (Canada): number analyzed (Participants) | 1292
  Month 26 - SF36 MH (Canada) | 81.76 (15.452)
  Month 38 - SF36 PF (Canada): number analyzed (Participants) | 1251
  Month 38 - SF36 PF (Canada) | 71.54 (25.455)
  Month 38 - SF36 RP (Canada): number analyzed (Participants) | 1252
  Month 38 - SF36 RP (Canada) | 75.04 (26.340)
  Month 38 - SF36 BP (Canada): number analyzed (Participants) | 1251
  Month 38 - SF36 BP (Canada) | 69.93 (24.498)
  Month 38 - SF36 GH (Canada): number analyzed (Participants) | 1252
  Month 38 - SF36 GH (Canada) | 73.81 (18.686)
  Month 38 - SF36 VT (Canada): number analyzed (Participants) | 1251
  Month 38 - SF36 VT (Canada) | 66.63 (19.059)
  Month 38 - SF36 SF (Canada): number analyzed (Participants) | 1251
  Month 38 - SF36 SF (Canada) | 85.69 (20.937)
  Month 38 - SF36 RE (Canada): number analyzed (Participants) | 1252
  Month 38 - SF36 RE (Canada) | 84.74 (22.316)
  Month 38 - SF36 MH (Canada): number analyzed (Participants) | 1251
  Month 38 - SF36 MH (Canada) | 80.52 (16.659)
  Month 0 - SF36 PF (Czechia): number analyzed (Participants) | 1226
  Month 0 - SF36 PF (Czechia) | 83.63 (16.758)
  Month 0 - SF36 RP (Czechia): number analyzed (Participants) | 1226
  Month 0 - SF36 RP (Czechia) | 83.52 (20.371)
  Month 0 - SF36 BP (Czechia): number analyzed (Participants) | 1226
  Month 0 - SF36 BP (Czechia) | 80.72 (23.278)
  Month 0 - SF36 GH (Czechia): number analyzed (Participants) | 1226
  Month 0 - SF36 GH (Czechia) | 68.85 (18.579)
  Month 0 - SF36 VT (Czechia): number analyzed (Participants) | 1226
  Month 0 - SF36 VT (Czechia) | 70.20 (17.658)
  Month 0 - SF36 SF (Czechia): number analyzed (Participants) | 1226
  Month 0 - SF36 SF (Czechia) | 89.77 (17.686)
  Month 0 - SF36 RE (Czechia): number analyzed (Participants) | 1226
  Month 0 - SF36 RE (Czechia) | 87.35 (18.853)
  Month 0 - SF36 MH (Czechia): number analyzed (Participants) | 1226
  Month 0 - SF36 MH (Czechia) | 78.85 (15.813)
  Month 14 - SF36 PF (Czechia): number analyzed (Participants) | 1210
  Month 14 - SF36 PF (Czechia) | 81.04 (20.182)
  Month 14 - SF36 RP (Czechia): number analyzed (Participants) | 1210
  Month 14 - SF36 RP (Czechia) | 71.82 (23.074)
  Month 14 - SF36 BP (Czechia): number analyzed (Participants) | 1210
  Month 14 - SF36 BP (Czechia) | 76.22 (25.263)
  Month 14 - SF36 GH (Czechia): number analyzed (Participants) | 1210
  Month 14 - SF36 GH (Czechia) | 67.28 (19.827)
  Month 14 - SF36 VT (Czechia): number analyzed (Participants) | 1210
  Month 14 - SF36 VT (Czechia) | 65.33 (18.155)
  Month 14 - SF36 SF (Czechia): number analyzed (Participants) | 1210
  Month 14 - SF36 SF (Czechia) | 84.17 (21.684)
  Month 14 - SF36 RE (Czechia): number analyzed (Participants) | 1210
  Month 14 - SF36 RE (Czechia) | 78.21 (21.121)
  Month 14 - SF36 MH (Czechia): number analyzed (Participants) | 1210
  Month 14 - SF36 MH (Czechia) | 74.13 (17.039)
  Month 26 - SF36 PF (Czechia): number analyzed (Participants) | 1199
  Month 26 - SF36 PF (Czechia) | 78.01 (22.368)
  Month 26 - SF36 RP (Czechia): number analyzed (Participants) | 1199
  Month 26 - SF36 RP (Czechia) | 68.18 (22.493)
  Month 26 - SF36 BP (Czechia): number analyzed (Participants) | 1199
  Month 26 - SF36 BP (Czechia) | 72.86 (25.494)
  Month 26 - SF36 GH (Czechia): number analyzed (Participants) | 1199
  Month 26 - SF36 GH (Czechia) | 64.08 (20.318)
  Month 26 - SF36 VT (Czechia): number analyzed (Participants) | 1199
  Month 26 - SF36 VT (Czechia) | 62.35 (18.222)
  Month 26 - SF36 SF (Czechia): number analyzed (Participants) | 1199
  Month 26 - SF36 SF (Czechia) | 81.68 (22.531)
  Month 26 - SF36 RE (Czechia): number analyzed (Participants) | 1199
  Month 26 - SF36 RE (Czechia) | 75.93 (22.099)
  Month 26 - SF36 MH (Czechia): number analyzed (Participants) | 1199
  Month 26 - SF36 MH (Czechia) | 72.47 (16.970)
  Month 38 - SF36 PF (Czechia): number analyzed (Participants) | 1177
  Month 38 - SF36 PF (Czechia) | 77.48 (22.752)
  Month 38 - SF36 RP (Czechia): number analyzed (Participants) | 1177
  Month 38 - SF36 RP (Czechia) | 67.50 (22.564)
  Month 38 - SF36 BP (Czechia): number analyzed (Participants) | 1177
  Month 38 - SF36 BP (Czechia) | 72.07 (25.893)
  Month 38 - SF36 GH (Czechia): number analyzed (Participants) | 1177
  Month 38 - SF36 GH (Czechia) | 64.39 (20.053)
  Month 38 - SF36 VT (Czechia): number analyzed (Participants) | 1177
  Month 38 - SF36 VT (Czechia) | 63.60 (17.688)
  Month 38 - SF36 SF (Czechia): number analyzed (Participants) | 1177
  Month 38 - SF36 SF (Czechia) | 82.13 (22.341)
  Month 38 - SF36 RE (Czechia): number analyzed (Participants) | 1177
  Month 38 - SF36 RE (Czechia) | 74.77 (22.306)
  Month 38 - SF36 MH (Czechia): number analyzed (Participants) | 1177
  Month 38 - SF36 MH (Czechia) | 72.78 (16.972)
  Month 0 - SF36 PF (Estonia): number analyzed (Participants) | 2125
  Month 0 - SF36 PF (Estonia) | 83.27 (18.040)
  Month 0 - SF36 RP (Estonia): number analyzed (Participants) | 2125
  Month 0 - SF36 RP (Estonia) | 77.52 (26.681)
  Month 0 - SF36 BP (Estonia): number analyzed (Participants) | 2125
  Month 0 - SF36 BP (Estonia) | 74.30 (24.729)
  Month 0 - SF36 GH (Estonia): number analyzed (Participants) | 2125
  Month 0 - SF36 GH (Estonia) | 58.49 (19.050)
  Month 0 - SF36 VT (Estonia): number analyzed (Participants) | 2125
  Month 0 - SF36 VT (Estonia) | 74.72 (17.041)
  Month 0 - SF36 SF (Estonia): number analyzed (Participants) | 2125
  Month 0 - SF36 SF (Estonia) | 91.78 (15.802)
  Month 0 - SF36 RE (Estonia): number analyzed (Participants) | 2125
  Month 0 - SF36 RE (Estonia) | 91.69 (16.141)
  Month 0 - SF36 MH (Estonia): number analyzed (Participants) | 2125
  Month 0 - SF36 MH (Estonia) | 80.04 (15.286)
  Month 14 - SF36 PF (Estonia): number analyzed (Participants) | 2059
  Month 14 - SF36 PF (Estonia) | 75.97 (23.487)
  Month 14 - SF36 RP (Estonia): number analyzed (Participants) | 2059
  Month 14 - SF36 RP (Estonia) | 77.40 (25.983)
  Month 14 - SF36 BP (Estonia): number analyzed (Participants) | 2059
  Month 14 - SF36 BP (Estonia) | 71.82 (25.076)
  Month 14 - SF36 GH (Estonia): number analyzed (Participants) | 2059
  Month 14 - SF36 GH (Estonia) | 57.17 (18.677)
  Month 14 - SF36 VT (Estonia): number analyzed (Participants) | 2059
  Month 14 - SF36 VT (Estonia) | 70.91 (18.447)
  Month 14 - SF36 SF (Estonia): number analyzed (Participants) | 2059
  Month 14 - SF36 SF (Estonia) | 91.00 (16.763)
  Month 14 - SF36 RE (Estonia): number analyzed (Participants) | 2059
  Month 14 - SF36 RE (Estonia) | 86.16 (21.264)
  Month 14 - SF36 MH (Estonia): number analyzed (Participants) | 2059
  Month 14 - SF36 MH (Estonia) | 79.17 (16.572)
  Month 26 - SF36 PF (Estonia): number analyzed (Participants) | 2031
  Month 26 - SF36 PF (Estonia) | 65.95 (26.066)
  Month 26 - SF36 RP (Estonia): number analyzed (Participants) | 2030
  Month 26 - SF36 RP (Estonia) | 67.55 (27.894)
  Month 26 - SF36 BP (Estonia): number analyzed (Participants) | 2030
  Month 26 - SF36 BP (Estonia) | 66.18 (25.194)
  Month 26 - SF36 GH (Estonia): number analyzed (Participants) | 2032
  Month 26 - SF36 GH (Estonia) | 52.15 (18.654)
  Month 26 - SF36 VT (Estonia): number analyzed (Participants) | 2031
  Month 26 - SF36 VT (Estonia) | 64.66 (19.248)
  Month 26 - SF36 SF (Estonia): number analyzed (Participants) | 2032
  Month 26 - SF36 SF (Estonia) | 84.31 (21.233)
  Month 26 - SF36 RE (Estonia): number analyzed (Participants) | 2030
  Month 26 - SF36 RE (Estonia) | 74.48 (26.156)
  Month 26 - SF36 MH (Estonia): number analyzed (Participants) | 2031
  Month 26 - SF36 MH (Estonia) | 74.94 (17.531)
  Month 38 - SF36 PF (Estonia): number analyzed (Participants) | 1994
  Month 38 - SF36 PF (Estonia) | 60.37 (26.153)
  Month 38 - SF36 RP (Estonia): number analyzed (Participants) | 1993
  Month 38 - SF36 RP (Estonia) | 62.11 (27.161)
  Month 38 - SF36 BP (Estonia): number analyzed (Participants) | 1994
  Month 38 - SF36 BP (Estonia) | 59.45 (23.335)
  Month 38 - SF36 GH (Estonia): number analyzed (Participants) | 1994
  Month 38 - SF36 GH (Estonia) | 48.53 (17.687)
  Month 38 - SF36 VT (Estonia): number analyzed (Participants) | 1994
  Month 38 - SF36 VT (Estonia) | 61.79 (18.816)
  Month 38 - SF36 SF (Estonia): number analyzed (Participants) | 1993
  Month 38 - SF36 SF (Estonia) | 81.45 (21.281)
  Month 38 - SF36 RE (Estonia): number analyzed (Participants) | 1993
  Month 38 - SF36 RE (Estonia) | 70.20 (26.084)
  Month 38 - SF36 MH (Estonia): number analyzed (Participants) | 1994
  Month 38 - SF36 MH (Estonia) | 73.08 (17.225)
  Month 0 - SF36 PF (Finland): number analyzed (Participants) | 3086
  Month 0 - SF36 PF (Finland) | 84.66 (17.428)
  Month 0 - SF36 RP (Finland): number analyzed (Participants) | 3088
  Month 0 - SF36 RP (Finland) | 86.35 (20.421)
  Month 0 - SF36 BP (Finland): number analyzed (Participants) | 3086
  Month 0 - SF36 BP (Finland) | 78.31 (20.019)
  Month 0 - SF36 GH (Finland): number analyzed (Participants) | 3113
  Month 0 - SF36 GH (Finland) | 72.29 (16.823)
  Month 0 - SF36 VT (Finland): number analyzed (Participants) | 3081
  Month 0 - SF36 VT (Finland) | 74.18 (16.187)
  Month 0 - SF36 SF (Finland): number analyzed (Participants) | 3103
  Month 0 - SF36 SF (Finland) | 94.09 (13.016)
  Month 0 - SF36 RE (Finland): number analyzed (Participants) | 3082
  Month 0 - SF36 RE (Finland) | 90.11 (17.475)
  Month 0 - SF36 MH (Finland): number analyzed (Participants) | 3079
  Month 0 - SF36 MH (Finland) | 86.54 (12.558)
  Month 14 - SF36 PF (Finland): number analyzed (Participants) | 2962
  Month 14 - SF36 PF (Finland) | 81.56 (20.057)
  Month 14 - SF36 RP (Finland): number analyzed (Participants) | 2964
  Month 14 - SF36 RP (Finland) | 82.89 (23.143)
  Month 14 - SF36 BP (Finland): number analyzed (Participants) | 2966
  Month 14 - SF36 BP (Finland) | 73.76 (22.297)
  Month 14 - SF36 GH (Finland): number analyzed (Participants) | 2979
  Month 14 - SF36 GH (Finland) | 69.35 (18.022)
  Month 14 - SF36 VT (Finland): number analyzed (Participants) | 2959
  Month 14 - SF36 VT (Finland) | 70.90 (18.617)
  Month 14 - SF36 SF (Finland): number analyzed (Participants) | 2976
  Month 14 - SF36 SF (Finland) | 91.98 (16.306)
  Month 14 - SF36 RE (Finland): number analyzed (Participants) | 2964
  Month 14 - SF36 RE (Finland) | 87.91 (19.929)
  Month 14 - SF36 MH (Finland): number analyzed (Participants) | 2960
  Month 14 - SF36 MH (Finland) | 85.49 (13.528)
  Month 26 - SF36 PF (Finland): number analyzed (Participants) | 2890
  Month 26 - SF36 PF (Finland) | 80.68 (20.609)
  Month 26 - SF36 RP (Finland): number analyzed (Participants) | 2891
  Month 26 - SF36 RP (Finland) | 81.29 (24.688)
  Month 26 - SF36 BP (Finland): number analyzed (Participants) | 2880
  Month 26 - SF36 BP (Finland) | 73.70 (22.313)
  Month 26 - SF36 GH (Finland): number analyzed (Participants) | 2903
  Month 26 - SF36 GH (Finland) | 68.25 (18.451)
  Month 26 - SF36 VT (Finland): number analyzed (Participants) | 2887
  Month 26 - SF36 VT (Finland) | 70.28 (18.764)
  Month 26 - SF36 SF (Finland): number analyzed (Participants) | 2900
  Month 26 - SF36 SF (Finland) | 91.13 (16.940)
  Month 26 - SF36 RE (Finland): number analyzed (Participants) | 2888
  Month 26 - SF36 RE (Finland) | 86.78 (20.806)
  Month 26 - SF36 MH (Finland): number analyzed (Participants) | 2887
  Month 26 - SF36 MH (Finland) | 84.90 (14.261)
  Month 38 - SF36 PF (Finland): number analyzed (Participants) | 2844
  Month 38 - SF36 PF (Finland) | 79.14 (21.864)
  Month 38 - SF36 RP (Finland): number analyzed (Participants) | 2850
  Month 38 - SF36 RP (Finland) | 79.86 (24.883)
  Month 38 - SF36 BP (Finland): number analyzed (Participants) | 2859
  Month 38 - SF36 BP (Finland) | 72.46 (22.635)
  Month 38 - SF36 GH (Finland): number analyzed (Participants) | 2864
  Month 38 - SF36 GH (Finland) | 66.89 (18.987)
  Month 38 - SF36 VT (Finland): number analyzed (Participants) | 2854
  Month 38 - SF36 VT (Finland) | 69.30 (19.226)
  Month 38 - SF36 SF (Finland): number analyzed (Participants) | 2864
  Month 38 - SF36 SF (Finland) | 90.65 (17.284)
  Month 38 - SF36 RE (Finland): number analyzed (Participants) | 2848
  Month 38 - SF36 RE (Finland) | 85.90 (21.204)
  Month 38 - SF36 MH (Finland): number analyzed (Participants) | 2854
  Month 38 - SF36 MH (Finland) | 84.54 (14.481)
  Month 0 - SF36 PF (France): number analyzed (Participants) | 1120
  Month 0 - SF36 PF (France) | 75.41 (24.712)
  Month 0 - SF36 RP (France): number analyzed (Participants) | 1121
  Month 0 - SF36 RP (France) | 73.50 (24.831)
  Month 0 - SF36 BP (France): number analyzed (Participants) | 1117
  Month 0 - SF36 BP (France) | 67.29 (23.946)
  Month 0 - SF36 GH (France): number analyzed (Participants) | 1121
  Month 0 - SF36 GH (France) | 64.74 (16.392)
  Month 0 - SF36 VT (France): number analyzed (Participants) | 1109
  Month 0 - SF36 VT (France) | 60.73 (18.170)
  Month 0 - SF36 SF (France): number analyzed (Participants) | 1117
  Month 0 - SF36 SF (France) | 80.61 (20.116)
  Month 0 - SF36 RE (France): number analyzed (Participants) | 1120
  Month 0 - SF36 RE (France) | 76.24 (24.041)
  Month 0 - SF36 MH (France): number analyzed (Participants) | 1110
  Month 0 - SF36 MH (France) | 67.97 (18.216)
  Month 14 - SF36 PF (France): number analyzed (Participants) | 1089
  Month 14 - SF36 PF (France) | 75.18 (24.455)
  Month 14 - SF36 RP (France): number analyzed (Participants) | 1087
  Month 14 - SF36 RP (France) | 70.95 (24.437)
  Month 14 - SF36 BP (France): number analyzed (Participants) | 1089
  Month 14 - SF36 BP (France) | 64.73 (23.409)
  Month 14 - SF36 GH (France): number analyzed (Participants) | 1091
  Month 14 - SF36 GH (France) | 62.80 (16.748)
  Month 14 - SF36 VT (France): number analyzed (Participants) | 1084
  Month 14 - SF36 VT (France) | 58.70 (18.280)
  Month 14 - SF36 SF (France): number analyzed (Participants) | 1090
  Month 14 - SF36 SF (France) | 76.55 (20.693)
  Month 14 - SF36 RE (France): number analyzed (Participants) | 1085
  Month 14 - SF36 RE (France) | 73.38 (23.899)
  Month 14 - SF36 MH (France): number analyzed (Participants) | 1083
  Month 14 - SF36 MH (France) | 66.77 (18.228)
  Month 26 - SF36 PF (France): number analyzed (Participants) | 1009
  Month 26 - SF36 PF (France) | 74.36 (24.684)
  Month 26 - SF36 RP (France): number analyzed (Participants) | 1012
  Month 26 - SF36 RP (France) | 68.23 (25.003)
  Month 26 - SF36 BP (France): number analyzed (Participants) | 1005
  Month 26 - SF36 BP (France) | 62.76 (23.949)
  Month 26 - SF36 GH (France): number analyzed (Participants) | 1014
  Month 26 - SF36 GH (France) | 61.46 (17.457)
  Month 26 - SF36 VT (France): number analyzed (Participants) | 1006
  Month 26 - SF36 VT (France) | 57.15 (19.107)
  Month 26 - SF36 SF (France): number analyzed (Participants) | 1009
  Month 26 - SF36 SF (France) | 74.86 (21.775)
  Month 26 - SF36 RE (France): number analyzed (Participants) | 1012
  Month 26 - SF36 RE (France) | 71.27 (24.405)
  Month 26 - SF36 MH (France): number analyzed (Participants) | 1006
  Month 26 - SF36 MH (France) | 65.37 (18.671)
  Month 38 - SF36 PF (France): number analyzed (Participants) | 996
  Month 38 - SF36 PF (France) | 74.03 (24.824)
  Month 38 - SF36 RP (France): number analyzed (Participants) | 995
  Month 38 - SF36 RP (France) | 67.99 (25.099)
  Month 38 - SF36 BP (France): number analyzed (Participants) | 995
  Month 38 - SF36 BP (France) | 62.02 (22.966)
  Month 38 - SF36 GH (France): number analyzed (Participants) | 997
  Month 38 - SF36 GH (France) | 60.60 (17.031)
  Month 38 - SF36 VT (France): number analyzed (Participants) | 993
  Month 38 - SF36 VT (France) | 56.85 (18.659)
  Month 38 - SF36 SF (France): number analyzed (Participants) | 997
  Month 38 - SF36 SF (France) | 73.68 (21.831)
  Month 38 - SF36 RE (France): number analyzed (Participants) | 996
  Month 38 - SF36 RE (France) | 71.29 (24.172)
  Month 38 - SF36 MH (France): number analyzed (Participants) | 993
  Month 38 - SF36 MH (France) | 65.49 (18.203)
  Month 0 - SF36 PF (Germany): number analyzed (Participants) | 1915
  Month 0 - SF36 PF (Germany) | 74.28 (24.865)
  Month 0 - SF36 RP (Germany): number analyzed (Participants) | 1919
  Month 0 - SF36 RP (Germany) | 72.36 (26.307)
  Month 0 - SF36 BP (Germany): number analyzed (Participants) | 1920
  Month 0 - SF36 BP (Germany) | 71.81 (27.520)
  Month 0 - SF36 GH (Germany): number analyzed (Participants) | 1921
  Month 0 - SF36 GH (Germany) | 67.79 (17.909)
  Month 0 - SF36 VT (Germany): number analyzed (Participants) | 1918
  Month 0 - SF36 VT (Germany) | 66.06 (18.835)
  Month 0 - SF36 SF (Germany): number analyzed (Participants) | 1920
  Month 0 - SF36 SF (Germany) | 87.35 (19.367)
  Month 0 - SF36 RE (Germany): number analyzed (Participants) | 1918
  Month 0 - SF36 RE (Germany) | 80.80 (24.970)
  Month 0 - SF36 MH (Germany): number analyzed (Participants) | 1918
  Month 0 - SF36 MH (Germany) | 76.40 (17.804)
  Month 14 - SF36 PF (Germany): number analyzed (Participants) | 1792
  Month 14 - SF36 PF (Germany) | 70.55 (26.402)
  Month 14 - SF36 RP (Germany): number analyzed (Participants) | 1817
  Month 14 - SF36 RP (Germany) | 70.53 (27.114)
  Month 14 - SF36 BP (Germany): number analyzed (Participants) | 1815
  Month 14 - SF36 BP (Germany) | 68.40 (28.031)
  Month 14 - SF36 GH (Germany): number analyzed (Participants) | 1818
  Month 14 - SF36 GH (Germany) | 65.86 (18.435)
  Month 14 - SF36 VT (Germany): number analyzed (Participants) | 1814
  Month 14 - SF36 VT (Germany) | 64.07 (19.605)
  Month 14 - SF36 SF (Germany): number analyzed (Participants) | 1817
  Month 14 - SF36 SF (Germany) | 86.44 (21.019)
  Month 14 - SF36 RE (Germany): number analyzed (Participants) | 1816
  Month 14 - SF36 RE (Germany) | 78.88 (26.001)
  Month 14 - SF36 MH (Germany): number analyzed (Participants) | 1814
  Month 14 - SF36 MH (Germany) | 75.30 (18.230)
  Month 26 - SF36 PF (Germany): number analyzed (Participants) | 1769
  Month 26 - SF36 PF (Germany) | 69.01 (26.633)
  Month 26 - SF36 RP (Germany): number analyzed (Participants) | 1771
  Month 26 - SF36 RP (Germany) | 67.97 (27.948)
  Month 26 - SF36 BP (Germany): number analyzed (Participants) | 1771
  Month 26 - SF36 BP (Germany) | 66.77 (28.555)
  Month 26 - SF36 GH (Germany): number analyzed (Participants) | 1773
  Month 26 - SF36 GH (Germany) | 64.65 (18.682)
  Month 26 - SF36 VT (Germany): number analyzed (Participants) | 1770
  Month 26 - SF36 VT (Germany) | 62.50 (19.903)
  Month 26 - SF36 SF (Germany): number analyzed (Participants) | 1773
  Month 26 - SF36 SF (Germany) | 84.84 (21.200)
  Month 26 - SF36 RE (Germany): number analyzed (Participants) | 1772
  Month 26 - SF36 RE (Germany) | 77.77 (26.354)
  Month 26 - SF36 MH (Germany): number analyzed (Participants) | 1769
  Month 26 - SF36 MH (Germany) | 74.49 (18.575)
  Month 38 - SF36 PF (Germany): number analyzed (Participants) | 1704
  Month 38 - SF36 PF (Germany) | 66.53 (27.718)
  Month 38 - SF36 RP (Germany): number analyzed (Participants) | 1702
  Month 38 - SF36 RP (Germany) | 65.12 (28.052)
  Month 38 - SF36 BP (Germany): number analyzed (Participants) | 1702
  Month 38 - SF36 BP (Germany) | 64.79 (28.435)
  Month 38 - SF36 GH (Germany): number analyzed (Participants) | 1704
  Month 38 - SF36 GH (Germany) | 62.92 (19.191)
  Month 38 - SF36 VT (Germany): number analyzed (Participants) | 1701
  Month 38 - SF36 VT (Germany) | 60.45 (20.033)
  Month 38 - SF36 SF (Germany): number analyzed (Participants) | 1704
  Month 38 - SF36 SF (Germany) | 82.56 (23.166)
  Month 38 - SF36 RE (Germany): number analyzed (Participants) | 1700
  Month 38 - SF36 RE (Germany) | 75.57 (26.996)
  Month 38 - SF36 MH (Germany): number analyzed (Participants) | 1701
  Month 38 - SF36 MH (Germany) | 72.80 (18.705)
  Month 0 - SF36 PF (Hong Kong): number analyzed (Participants) | 648
  Month 0 - SF36 PF (Hong Kong) | 83.21 (18.057)
  Month 0 - SF36 RP (Hong Kong): number analyzed (Participants) | 648
  Month 0 - SF36 RP (Hong Kong) | 80.34 (21.511)
  Month 0 - SF36 BP (Hong Kong): number analyzed (Participants) | 648
  Month 0 - SF36 BP (Hong Kong) | 70.96 (23.972)
  Month 0 - SF36 GH (Hong Kong): number analyzed (Participants) | 648
  Month 0 - SF36 GH (Hong Kong) | 64.98 (18.295)
  Month 0 - SF36 VT (Hong Kong): number analyzed (Participants) | 647
  Month 0 - SF36 VT (Hong Kong) | 67.55 (18.230)
  Month 0 - SF36 SF (Hong Kong): number analyzed (Participants) | 648
  Month 0 - SF36 SF (Hong Kong) | 85.80 (18.176)
  Month 0 - SF36 RE (Hong Kong): number analyzed (Participants) | 648
  Month 0 - SF36 RE (Hong Kong) | 82.16 (19.210)
  Month 0 - SF36 MH (Hong Kong): number analyzed (Participants) | 647
  Month 0 - SF36 MH (Hong Kong) | 75.43 (16.891)
  Month 14 - SF36 PF (Hong Kong): number analyzed (Participants) | 622
  Month 14 - SF36 PF (Hong Kong) | 79.35 (20.242)
  Month 14 - SF36 RP (Hong Kong): number analyzed (Participants) | 622
  Month 14 - SF36 RP (Hong Kong) | 75.11 (23.850)
  Month 14 - SF36 BP (Hong Kong): number analyzed (Participants) | 622
  Month 14 - SF36 BP (Hong Kong) | 67.98 (24.349)
  Month 14 - SF36 GH (Hong Kong): number analyzed (Participants) | 622
  Month 14 - SF36 GH (Hong Kong) | 62.23 (19.396)
  Month 14 - SF36 VT (Hong Kong): number analyzed (Participants) | 622
  Month 14 - SF36 VT (Hong Kong) | 64.27 (19.121)
  Month 14 - SF36 SF (Hong Kong): number analyzed (Participants) | 622
  Month 14 - SF36 SF (Hong Kong) | 81.83 (21.223)
  Month 14 - SF36 RE (Hong Kong): number analyzed (Participants) | 622
  Month 14 - SF36 RE (Hong Kong) | 77.99 (22.505)
  Month 14 - SF36 MH (Hong Kong): number analyzed (Participants) | 622
  Month 14 - SF36 MH (Hong Kong) | 73.79 (17.471)
  Month 26 - SF36 PF (Hong Kong): number analyzed (Participants) | 604
  Month 26 - SF36 PF (Hong Kong) | 78.42 (21.721)
  Month 26 - SF36 RP (Hong Kong): number analyzed (Participants) | 604
  Month 26 - SF36 RP (Hong Kong) | 75.63 (24.198)
  Month 26 - SF36 BP (Hong Kong): number analyzed (Participants) | 604
  Month 26 - SF36 BP (Hong Kong) | 68.43 (23.730)
  Month 26 - SF36 GH (Hong Kong): number analyzed (Participants) | 604
  Month 26 - SF36 GH (Hong Kong) | 61.23 (20.163)
  Month 26 - SF36 VT (Hong Kong): number analyzed (Participants) | 604
  Month 26 - SF36 VT (Hong Kong) | 63.51 (19.771)
  Month 26 - SF36 SF (Hong Kong): number analyzed (Participants) | 604
  Month 26 - SF36 SF (Hong Kong) | 80.96 (21.922)
  Month 26 - SF36 RE (Hong Kong): number analyzed (Participants) | 604
  Month 26 - SF36 RE (Hong Kong) | 77.75 (23.055)
  Month 26 - SF36 MH (Hong Kong): number analyzed (Participants) | 604
  Month 26 - SF36 MH (Hong Kong) | 73.15 (16.489)
  Month 38 - SF36 PF (Hong Kong): number analyzed (Participants) | 595
  Month 38 - SF36 PF (Hong Kong) | 77.54 (22.833)
  Month 38 - SF36 RP (Hong Kong): number analyzed (Participants) | 595
  Month 38 - SF36 RP (Hong Kong) | 73.67 (24.805)
  Month 38 - SF36 BP (Hong Kong): number analyzed (Participants) | 595
  Month 38 - SF36 BP (Hong Kong) | 67.34 (24.483)
  Month 38 - SF36 GH (Hong Kong): number analyzed (Participants) | 595
  Month 38 - SF36 GH (Hong Kong) | 61.39 (19.740)
  Month 38 - SF36 VT (Hong Kong): number analyzed (Participants) | 595
  Month 38 - SF36 VT (Hong Kong) | 64.05 (20.721)
  Month 38 - SF36 SF (Hong Kong): number analyzed (Participants) | 595
  Month 38 - SF36 SF (Hong Kong) | 81.62 (21.797)
  Month 38 - SF36 RE (Hong Kong): number analyzed (Participants) | 595
  Month 38 - SF36 RE (Hong Kong) | 76.32 (24.373)
  Month 38 - SF36 MH (Hong Kong): number analyzed (Participants) | 595
  Month 38 - SF36 MH (Hong Kong) | 72.82 (17.329)
  Month 0 - SF36 PF (Italy): number analyzed (Participants) | 278
  Month 0 - SF36 PF (Italy) | 86.53 (19.730)
  Month 0 - SF36 RP (Italy): number analyzed (Participants) | 277
  Month 0 - SF36 RP (Italy) | 82.24 (23.022)
  Month 0 - SF36 BP (Italy): number analyzed (Participants) | 278
  Month 0 - SF36 BP (Italy) | 77.60 (22.612)
  Month 0 - SF36 GH (Italy): number analyzed (Participants) | 278
  Month 0 - SF36 GH (Italy) | 68.83 (16.936)
  Month 0 - SF36 VT (Italy): number analyzed (Participants) | 278
  Month 0 - SF36 VT (Italy) | 69.02 (16.438)
  Month 0 - SF36 SF (Italy): number analyzed (Participants) | 278
  Month 0 - SF36 SF (Italy) | 83.32 (18.086)
  Month 0 - SF36 RE (Italy): number analyzed (Participants) | 277
  Month 0 - SF36 RE (Italy) | 81.83 (23.533)
  Month 0 - SF36 MH (Italy): number analyzed (Participants) | 278
  Month 0 - SF36 MH (Italy) | 74.33 (16.931)
  Month 14 - SF36 PF (Italy): number analyzed (Participants) | 264
  Month 14 - SF36 PF (Italy) | 87.31 (15.749)
  Month 14 - SF36 RP (Italy): number analyzed (Participants) | 264
  Month 14 - SF36 RP (Italy) | 80.85 (22.119)
  Month 14 - SF36 BP (Italy): number analyzed (Participants) | 263
  Month 14 - SF36 BP (Italy) | 76.25 (23.474)
  Month 14 - SF36 GH (Italy): number analyzed (Participants) | 264
  Month 14 - SF36 GH (Italy) | 67.43 (15.923)
  Month 14 - SF36 VT (Italy): number analyzed (Participants) | 264
  Month 14 - SF36 VT (Italy) | 67.05 (16.316)
  Month 14 - SF36 SF (Italy): number analyzed (Participants) | 264
  Month 14 - SF36 SF (Italy) | 82.81 (18.593)
  Month 14 - SF36 RE (Italy): number analyzed (Participants) | 264
  Month 14 - SF36 RE (Italy) | 83.11 (19.246)
  Month 14 - SF36 MH (Italy): number analyzed (Participants) | 264
  Month 14 - SF36 MH (Italy) | 73.56 (15.655)
  Month 26 - SF36 PF (Italy): number analyzed (Participants) | 251
  Month 26 - SF36 PF (Italy) | 86.19 (18.527)
  Month 26 - SF36 RP (Italy): number analyzed (Participants) | 251
  Month 26 - SF36 RP (Italy) | 79.01 (23.544)
  Month 26 - SF36 BP (Italy): number analyzed (Participants) | 251
  Month 26 - SF36 BP (Italy) | 74.54 (24.129)
  Month 26 - SF36 GH (Italy): number analyzed (Participants) | 251
  Month 26 - SF36 GH (Italy) | 65.89 (16.558)
  Month 26 - SF36 VT (Italy): number analyzed (Participants) | 251
  Month 26 - SF36 VT (Italy) | 66.65 (16.440)
  Month 26 - SF36 SF (Italy): number analyzed (Participants) | 251
  Month 26 - SF36 SF (Italy) | 80.43 (19.963)
  Month 26 - SF36 RE (Italy): number analyzed (Participants) | 251
  Month 26 - SF36 RE (Italy) | 82.50 (21.230)
  Month 26 - SF36 MH (Italy): number analyzed (Participants) | 251
  Month 26 - SF36 MH (Italy) | 72.73 (16.689)
  Month 38 - SF36 PF (Italy): number analyzed (Participants) | 243
  Month 38 - SF36 PF (Italy) | 84.73 (18.063)
  Month 38 - SF36 RP (Italy): number analyzed (Participants) | 243
  Month 38 - SF36 RP (Italy) | 77.37 (23.479)
  Month 38 - SF36 BP (Italy): number analyzed (Participants) | 242
  Month 38 - SF36 BP (Italy) | 73.01 (23.983)
  Month 38 - SF36 GH (Italy): number analyzed (Participants) | 243
  Month 38 - SF36 GH (Italy) | 63.52 (17.528)
  Month 38 - SF36 VT (Italy): number analyzed (Participants) | 240
  Month 38 - SF36 VT (Italy) | 63.63 (18.488)
  Month 38 - SF36 SF (Italy): number analyzed (Participants) | 242
  Month 38 - SF36 SF (Italy) | 78.82 (20.455)
  Month 38 - SF36 RE (Italy): number analyzed (Participants) | 242
  Month 38 - SF36 RE (Italy) | 79.55 (22.863)
  Month 38 - SF36 MH (Italy): number analyzed (Participants) | 240
  Month 38 - SF36 MH (Italy) | 70.74 (17.479)
  Month 0 - SF36 PF (Japan): number analyzed (Participants) | 771
  Month 0 - SF36 PF (Japan) | 88.88 (12.908)
  Month 0 - SF36 RP (Japan): number analyzed (Participants) | 771
  Month 0 - SF36 RP (Japan) | 91.82 (16.302)
  Month 0 - SF36 BP (Japan): number analyzed (Participants) | 771
  Month 0 - SF36 BP (Japan) | 82.43 (19.448)
  Month 0 - SF36 GH (Japan): number analyzed (Participants) | 771
  Month 0 - SF36 GH (Japan) | 70.69 (15.760)
  Month 0 - SF36 VT (Japan): number analyzed (Participants) | 771
  Month 0 - SF36 VT (Japan) | 73.62 (17.006)
  Month 0 - SF36 SF (Japan): number analyzed (Participants) | 771
  Month 0 - SF36 SF (Japan) | 92.56 (14.706)
  Month 0 - SF36 RE (Japan): number analyzed (Participants) | 771
  Month 0 - SF36 RE (Japan) | 92.63 (15.595)
  Month 0 - SF36 MH (Japan): number analyzed (Participants) | 771
  Month 0 - SF36 MH (Japan) | 81.22 (15.266)
  Month 14 - SF36 PF (Japan): number analyzed (Participants) | 738
  Month 14 - SF36 PF (Japan) | 89.69 (12.128)
  Month 14 - SF36 RP (Japan): number analyzed (Participants) | 738
  Month 14 - SF36 RP (Japan) | 91.48 (17.297)
  Month 14 - SF36 BP (Japan): number analyzed (Participants) | 738
  Month 14 - SF36 BP (Japan) | 80.18 (21.763)
  Month 14 - SF36 GH (Japan): number analyzed (Participants) | 738
  Month 14 - SF36 GH (Japan) | 71.51 (16.647)
  Month 14 - SF36 VT (Japan): number analyzed (Participants) | 738
  Month 14 - SF36 VT (Japan) | 73.72 (18.533)
  Month 14 - SF36 SF (Japan): number analyzed (Participants) | 738
  Month 14 - SF36 SF (Japan) | 92.65 (15.728)
  Month 14 - SF36 RE (Japan): number analyzed (Participants) | 738
  Month 14 - SF36 RE (Japan) | 92.71 (15.618)
  Month 14 - SF36 MH (Japan): number analyzed (Participants) | 738
  Month 14 - SF36 MH (Japan) | 81.94 (16.363)
  Month 26 - SF36 PF (Japan): number analyzed (Participants) | 723
  Month 26 - SF36 PF (Japan) | 87.94 (14.652)
  Month 26 - SF36 RP (Japan): number analyzed (Participants) | 723
  Month 26 - SF36 RP (Japan) | 90.40 (18.839)
  Month 26 - SF36 BP (Japan): number analyzed (Participants) | 723
  Month 26 - SF36 BP (Japan) | 80.13 (20.899)
  Month 26 - SF36 GH (Japan): number analyzed (Participants) | 723
  Month 26 - SF36 GH (Japan) | 70.08 (17.053)
  Month 26 - SF36 VT (Japan): number analyzed (Participants) | 723
  Month 26 - SF36 VT (Japan) | 72.86 (18.257)
  Month 26 - SF36 SF (Japan): number analyzed (Participants) | 723
  Month 26 - SF36 SF (Japan) | 91.75 (16.104)
  Month 26 - SF36 RE (Japan): number analyzed (Participants) | 723
  Month 26 - SF36 RE (Japan) | 92.62 (15.921)
  Month 26 - SF36 MH (Japan): number analyzed (Participants) | 723
  Month 26 - SF36 MH (Japan) | 82.25 (15.763)
  Month 38 - SF36 PF (Japan): number analyzed (Participants) | 702
  Month 38 - SF36 PF (Japan) | 87.65 (16.327)
  Month 38 - SF36 RP (Japan): number analyzed (Participants) | 702
  Month 38 - SF36 RP (Japan) | 89.75 (19.328)
  Month 38 - SF36 BP (Japan): number analyzed (Participants) | 702
  Month 38 - SF36 BP (Japan) | 80.38 (21.386)
  Month 38 - SF36 GH (Japan): number analyzed (Participants) | 702
  Month 38 - SF36 GH (Japan) | 69.72 (17.798)
  Month 38 - SF36 VT (Japan): number analyzed (Participants) | 702
  Month 38 - SF36 VT (Japan) | 71.77 (19.749)
  Month 38 - SF36 SF (Japan): number analyzed (Participants) | 702
  Month 38 - SF36 SF (Japan) | 91.81 (16.776)
  Month 38 - SF36 RE (Japan): number analyzed (Participants) | 702
  Month 38 - SF36 RE (Japan) | 91.44 (17.817)
  Month 38 - SF36 MH (Japan): number analyzed (Participants) | 702
  Month 38 - SF36 MH (Japan) | 81.69 (16.549)
  Month 0 - SF36 PF (Republic of Korea): number analyzed (Participants) | 1066
  Month 0 - SF36 PF (Republic of Korea) | 67.77 (26.978)
  Month 0 - SF36 RP (Republic of Korea): number analyzed (Participants) | 1066
  Month 0 - SF36 RP (Republic of Korea) | 77.43 (28.253)
  Month 0 - SF36 BP (Republic of Korea): number analyzed (Participants) | 1066
  Month 0 - SF36 BP (Republic of Korea) | 77.21 (22.831)
  Month 0 - SF36 GH (Republic of Korea): number analyzed (Participants) | 1066
  Month 0 - SF36 GH (Republic of Korea) | 63.51 (17.871)
  Month 0 - SF36 VT (Republic of Korea): number analyzed (Participants) | 1066
  Month 0 - SF36 VT (Republic of Korea) | 62.41 (21.822)
  Month 0 - SF36 SF (Republic of Korea): number analyzed (Participants) | 1066
  Month 0 - SF36 SF (Republic of Korea) | 88.91 (18.000)
  Month 0 - SF36 RE (Republic of Korea): number analyzed (Participants) | 1066
  Month 0 - SF36 RE (Republic of Korea) | 82.90 (25.455)
  Month 0 - SF36 MH (Republic of Korea): number analyzed (Participants) | 1066
  Month 0 - SF36 MH (Republic of Korea) | 77.15 (17.804)
  Month 14 - SF36 PF (Republic of Korea): number analyzed (Participants) | 940
  Month 14 - SF36 PF (Republic of Korea) | 68.09 (25.214)
  Month 14 - SF36 RP (Republic of Korea): number analyzed (Participants) | 940
  Month 14 - SF36 RP (Republic of Korea) | 79.45 (27.205)
  Month 14 - SF36 BP (Republic of Korea): number analyzed (Participants) | 940
  Month 14 - SF36 BP (Republic of Korea) | 76.12 (23.543)
  Month 14 - SF36 GH (Republic of Korea): number analyzed (Participants) | 940
  Month 14 - SF36 GH (Republic of Korea) | 60.18 (17.724)
  Month 14 - SF36 VT (Republic of Korea): number analyzed (Participants) | 940
  Month 14 - SF36 VT (Republic of Korea) | 58.10 (22.111)
  Month 14 - SF36 SF (Republic of Korea): number analyzed (Participants) | 940
  Month 14 - SF36 SF (Republic of Korea) | 88.24 (19.223)
  Month 14 - SF36 RE (Republic of Korea): number analyzed (Participants) | 940
  Month 14 - SF36 RE (Republic of Korea) | 82.54 (25.203)
  Month 14 - SF36 MH (Republic of Korea): number analyzed (Participants) | 940
  Month 14 - SF36 MH (Republic of Korea) | 73.41 (19.630)
  Month 26 - SF36 PF (Republic of Korea): number analyzed (Participants) | 905
  Month 26 - SF36 PF (Republic of Korea) | 68.22 (27.279)
  Month 26 - SF36 RP (Republic of Korea): number analyzed (Participants) | 905
  Month 26 - SF36 RP (Republic of Korea) | 77.15 (29.110)
  Month 26 - SF36 BP (Republic of Korea): number analyzed (Participants) | 906
  Month 26 - SF36 BP (Republic of Korea) | 76.05 (22.808)
  Month 26 - SF36 GH (Republic of Korea): number analyzed (Participants) | 906
  Month 26 - SF36 GH (Republic of Korea) | 59.59 (17.585)
  Month 26 - SF36 VT (Republic of Korea): number analyzed (Participants) | 905
  Month 26 - SF36 VT (Republic of Korea) | 56.19 (20.988)
  Month 26 - SF36 SF (Republic of Korea): number analyzed (Participants) | 906
  Month 26 - SF36 SF (Republic of Korea) | 88.00 (18.962)
  Month 26 - SF36 RE (Republic of Korea): number analyzed (Participants) | 906
  Month 26 - SF36 RE (Republic of Korea) | 83.44 (24.461)
  Month 26 - SF36 MH (Republic of Korea): number analyzed (Participants) | 905
  Month 26 - SF36 MH (Republic of Korea) | 73.31 (18.120)
  Month 38 - SF36 PF (Republic of Korea): number analyzed (Participants) | 862
  Month 38 - SF36 PF (Republic of Korea) | 68.77 (24.394)
  Month 38 - SF36 RP (Republic of Korea): number analyzed (Participants) | 863
  Month 38 - SF36 RP (Republic of Korea) | 77.22 (28.780)
  Month 38 - SF36 BP (Republic of Korea): number analyzed (Participants) | 863
  Month 38 - SF36 BP (Republic of Korea) | 75.94 (23.169)
  Month 38 - SF36 GH (Republic of Korea): number analyzed (Participants) | 863
  Month 38 - SF36 GH (Republic of Korea) | 60.91 (18.678)
  Month 38 - SF36 VT (Republic of Korea): number analyzed (Participants) | 862
  Month 38 - SF36 VT (Republic of Korea) | 59.99 (21.325)
  Month 38 - SF36 SF (Republic of Korea): number analyzed (Participants) | 863
  Month 38 - SF36 SF (Republic of Korea) | 87.37 (20.181)
  Month 38 - SF36 RE (Republic of Korea): number analyzed (Participants) | 863
  Month 38 - SF36 RE (Republic of Korea) | 82.99 (24.826)
  Month 38 - SF36 MH (Republic of Korea): number analyzed (Participants) | 862
  Month 38 - SF36 MH (Republic of Korea) | 72.97 (18.246)
  Month 0 - SF36 PF (Mexico): number analyzed (Participants) | 928
  Month 0 - SF36 PF (Mexico) | 76.06 (24.708)
  Month 0 - SF36 RP (Mexico): number analyzed (Participants) | 928
  Month 0 - SF36 RP (Mexico) | 75.05 (25.724)
  Month 0 - SF36 BP (Mexico): number analyzed (Participants) | 929
  Month 0 - SF36 BP (Mexico) | 73.03 (24.251)
  Month 0 - SF36 GH (Mexico): number analyzed (Participants) | 929
  Month 0 - SF36 GH (Mexico) | 64.84 (21.693)
  Month 0 - SF36 VT (Mexico): number analyzed (Participants) | 929
  Month 0 - SF36 VT (Mexico) | 68.62 (19.869)
  Month 0 - SF36 SF (Mexico): number analyzed (Participants) | 929
  Month 0 - SF36 SF (Mexico) | 81.98 (20.943)
  Month 0 - SF36 RE (Mexico): number analyzed (Participants) | 928
  Month 0 - SF36 RE (Mexico) | 77.19 (23.958)
  Month 0 - SF36 MH (Mexico): number analyzed (Participants) | 929
  Month 0 - SF36 MH (Mexico) | 72.17 (19.691)
  Month 14 - SF36 PF (Mexico): number analyzed (Participants) | 818
  Month 14 - SF36 PF (Mexico) | 73.73 (25.765)
  Month 14 - SF36 RP (Mexico): number analyzed (Participants) | 819
  Month 14 - SF36 RP (Mexico) | 76.33 (28.535)
  Month 14 - SF36 BP (Mexico): number analyzed (Participants) | 819
  Month 14 - SF36 BP (Mexico) | 71.34 (27.257)
  Month 14 - SF36 GH (Mexico): number analyzed (Participants) | 819
  Month 14 - SF36 GH (Mexico) | 63.83 (24.663)
  Month 14 - SF36 VT (Mexico): number analyzed (Participants) | 819
  Month 14 - SF36 VT (Mexico) | 67.13 (23.573)
  Month 14 - SF36 SF (Mexico): number analyzed (Participants) | 819
  Month 14 - SF36 SF (Mexico) | 84.19 (23.017)
  Month 14 - SF36 RE (Mexico): number analyzed (Participants) | 819
  Month 14 - SF36 RE (Mexico) | 81.86 (25.777)
  Month 14 - SF36 MH (Mexico): number analyzed (Participants) | 819
  Month 14 - SF36 MH (Mexico) | 73.26 (22.822)
  Month 26 - SF36 PF (Mexico): number analyzed (Participants) | 785
  Month 26 - SF36 PF (Mexico) | 69.20 (27.709)
  Month 26 - SF36 RP (Mexico): number analyzed (Participants) | 785
  Month 26 - SF36 RP (Mexico) | 76.59 (27.985)
  Month 26 - SF36 BP (Mexico): number analyzed (Participants) | 785
  Month 26 - SF36 BP (Mexico) | 70.63 (26.378)
  Month 26 - SF36 GH (Mexico): number analyzed (Participants) | 785
  Month 26 - SF36 GH (Mexico) | 61.32 (24.274)
  Month 26 - SF36 VT (Mexico): number analyzed (Participants) | 785
  Month 26 - SF36 VT (Mexico) | 65.73 (24.304)
  Month 26 - SF36 SF (Mexico): number analyzed (Participants) | 785
  Month 26 - SF36 SF (Mexico) | 83.33 (22.879)
  Month 26 - SF36 RE (Mexico): number analyzed (Participants) | 785
  Month 26 - SF36 RE (Mexico) | 80.72 (25.848)
  Month 26 - SF36 MH (Mexico): number analyzed (Participants) | 785
  Month 26 - SF36 MH (Mexico) | 73.30 (22.825)
  Month 38 - SF36 PF (Mexico): number analyzed (Participants) | 749
  Month 38 - SF36 PF (Mexico) | 65.25 (28.863)
  Month 38 - SF36 RP (Mexico): number analyzed (Participants) | 749
  Month 38 - SF36 RP (Mexico) | 70.65 (29.950)
  Month 38 - SF36 BP (Mexico): number analyzed (Participants) | 749
  Month 38 - SF36 BP (Mexico) | 67.32 (26.220)
  Month 38 - SF36 GH (Mexico): number analyzed (Participants) | 749
  Month 38 - SF36 GH (Mexico) | 59.99 (23.909)
  Month 38 - SF36 VT (Mexico): number analyzed (Participants) | 749
  Month 38 - SF36 VT (Mexico) | 63.93 (23.206)
  Month 38 - SF36 SF (Mexico): number analyzed (Participants) | 749
  Month 38 - SF36 SF (Mexico) | 78.10 (25.405)
  Month 38 - SF36 RE (Mexico): number analyzed (Participants) | 749
  Month 38 - SF36 RE (Mexico) | 73.58 (28.335)
  Month 38 - SF36 MH (Mexico): number analyzed (Participants) | 749
  Month 38 - SF36 MH (Mexico) | 71.19 (21.882)
  Month 0 - SF36 PF (Spain): number analyzed (Participants) | 1986
  Month 0 - SF36 PF (Spain) | 79.28 (21.596)
  Month 0 - SF36 RP (Spain): number analyzed (Participants) | 1986
  Month 0 - SF36 RP (Spain) | 87.75 (21.338)
  Month 0 - SF36 BP (Spain): number analyzed (Participants) | 1987
  Month 0 - SF36 BP (Spain) | 76.05 (24.753)
  Month 0 - SF36 GH (Spain): number analyzed (Participants) | 1987
  Month 0 - SF36 GH (Spain) | 68.73 (18.313)
  Month 0 - SF36 VT (Spain): number analyzed (Participants) | 1987
  Month 0 - SF36 VT (Spain) | 74.00 (20.813)
  Month 0 - SF36 SF (Spain): number analyzed (Participants) | 1987
  Month 0 - SF36 SF (Spain) | 91.18 (17.192)
  Month 0 - SF36 RE (Spain): number analyzed (Participants) | 1986
  Month 0 - SF36 RE (Spain) | 91.34 (17.970)
  Month 0 - SF36 MH (Spain): number analyzed (Participants) | 1987
  Month 0 - SF36 MH (Spain) | 80.26 (19.405)
  Month 14 - SF36 PF (Spain): number analyzed (Participants) | 1850
  Month 14 - SF36 PF (Spain) | 75.49 (24.090)
  Month 14 - SF36 RP (Spain): number analyzed (Participants) | 1850
  Month 14 - SF36 RP (Spain) | 85.12 (23.307)
  Month 14 - SF36 BP (Spain): number analyzed (Participants) | 1849
  Month 14 - SF36 BP (Spain) | 71.39 (26.702)
  Month 14 - SF36 GH (Spain): number analyzed (Participants) | 1850
  Month 14 - SF36 GH (Spain) | 67.05 (19.516)
  Month 14 - SF36 VT (Spain): number analyzed (Participants) | 1848
  Month 14 - SF36 VT (Spain) | 68.42 (23.055)
  Month 14 - SF36 SF (Spain): number analyzed (Participants) | 1850
  Month 14 - SF36 SF (Spain) | 88.13 (21.275)
  Month 14 - SF36 RE (Spain): number analyzed (Participants) | 1850
  Month 14 - SF36 RE (Spain) | 89.69 (20.295)
  Month 14 - SF36 MH (Spain): number analyzed (Participants) | 1847
  Month 14 - SF36 MH (Spain) | 76.22 (20.698)
  Month 26 - SF36 PF (Spain): number analyzed (Participants) | 1795
  Month 26 - SF36 PF (Spain) | 74.18 (24.468)
  Month 26 - SF36 RP (Spain): number analyzed (Participants) | 1794
  Month 26 - SF36 RP (Spain) | 81.33 (26.181)
  Month 26 - SF36 BP (Spain): number analyzed (Participants) | 1795
  Month 26 - SF36 BP (Spain) | 69.64 (27.123)
  Month 26 - SF36 GH (Spain): number analyzed (Participants) | 1795
  Month 26 - SF36 GH (Spain) | 66.01 (19.368)
  Month 26 - SF36 VT (Spain): number analyzed (Participants) | 1793
  Month 26 - SF36 VT (Spain) | 66.97 (23.292)
  Month 26 - SF36 SF (Spain): number analyzed (Participants) | 1795
  Month 26 - SF36 SF (Spain) | 87.43 (21.646)
  Month 26 - SF36 RE (Spain): number analyzed (Participants) | 1794
  Month 26 - SF36 RE (Spain) | 88.43 (21.561)
  Month 26 - SF36 MH (Spain): number analyzed (Participants) | 1793
  Month 26 - SF36 MH (Spain) | 75.64 (20.759)
  Month 38 - SF36 PF (Spain): number analyzed (Participants) | 1744
  Month 38 - SF36 PF (Spain) | 72.59 (25.686)
  Month 38 - SF36 RP (Spain): number analyzed (Participants) | 1743
  Month 38 - SF36 RP (Spain) | 81.18 (26.008)
  Month 38 - SF36 BP (Spain): number analyzed (Participants) | 1743
  Month 38 - SF36 BP (Spain) | 69.62 (26.974)
  Month 38 - SF36 GH (Spain): number analyzed (Participants) | 1745
  Month 38 - SF36 GH (Spain) | 64.83 (19.604)
  Month 38 - SF36 VT (Spain): number analyzed (Participants) | 1743
  Month 38 - SF36 VT (Spain) | 65.44 (23.097)
  Month 38 - SF36 SF (Spain): number analyzed (Participants) | 1744
  Month 38 - SF36 SF (Spain) | 87.16 (21.780)
  Month 38 - SF36 RE (Spain): number analyzed (Participants) | 1742
  Month 38 - SF36 RE (Spain) | 88.97 (20.277)
  Month 38 - SF36 MH (Spain): number analyzed (Participants) | 1742
  Month 38 - SF36 MH (Spain) | 75.14 (20.731)
  Month 0 - SF36 PF (Sweden): number analyzed (Participants) | 1748
  Month 0 - SF36 PF (Sweden) | 84.11 (18.733)
  Month 0 - SF36 RP (Sweden): number analyzed (Participants) | 1747
  Month 0 - SF36 RP (Sweden) | 88.84 (19.401)
  Month 0 - SF36 BP (Sweden): number analyzed (Participants) | 1746
  Month 0 - SF36 BP (Sweden) | 79.07 (22.648)
  Month 0 - SF36 GH (Sweden): number analyzed (Participants) | 1753
  Month 0 - SF36 GH (Sweden) | 80.36 (17.091)
  Month 0 - SF36 VT (Sweden): number analyzed (Participants) | 1745
  Month 0 - SF36 VT (Sweden) | 76.15 (18.033)
  Month 0 - SF36 SF (Sweden): number analyzed (Participants) | 1747
  Month 0 - SF36 SF (Sweden) | 93.78 (14.547)
  Month 0 - SF36 RE (Sweden): number analyzed (Participants) | 1746
  Month 0 - SF36 RE (Sweden) | 92.59 (16.008)
  Month 0 - SF36 MH (Sweden): number analyzed (Participants) | 1745
  Month 0 - SF36 MH (Sweden) | 87.01 (13.481)
  Month 14 - SF36 PF (Sweden): number analyzed (Participants) | 1683
  Month 14 - SF36 PF (Sweden) | 81.48 (20.319)
  Month 14 - SF36 RP (Sweden): number analyzed (Participants) | 1682
  Month 14 - SF36 RP (Sweden) | 85.40 (22.576)
  Month 14 - SF36 BP (Sweden): number analyzed (Participants) | 1675
  Month 14 - SF36 BP (Sweden) | 75.90 (24.641)
  Month 14 - SF36 GH (Sweden): number analyzed (Participants) | 1684
  Month 14 - SF36 GH (Sweden) | 76.00 (18.800)
  Month 14 - SF36 VT (Sweden): number analyzed (Participants) | 1678
  Month 14 - SF36 VT (Sweden) | 73.01 (20.496)
  Month 14 - SF36 SF (Sweden): number analyzed (Participants) | 1678
  Month 14 - SF36 SF (Sweden) | 91.60 (17.418)
  Month 14 - SF36 RE (Sweden): number analyzed (Participants) | 1682
  Month 14 - SF36 RE (Sweden) | 90.96 (18.262)
  Month 14 - SF36 MH (Sweden): number analyzed (Participants) | 1678
  Month 14 - SF36 MH (Sweden) | 86.18 (14.848)
  Month 26 - SF36 PF (Sweden): number analyzed (Participants) | 1655
  Month 26 - SF36 PF (Sweden) | 80.67 (20.988)
  Month 26 - SF36 RP (Sweden): number analyzed (Participants) | 1656
  Month 26 - SF36 RP (Sweden) | 84.62 (23.270)
  Month 26 - SF36 BP (Sweden): number analyzed (Participants) | 1653
  Month 26 - SF36 BP (Sweden) | 75.01 (24.387)
  Month 26 - SF36 GH (Sweden): number analyzed (Participants) | 1659
  Month 26 - SF36 GH (Sweden) | 75.90 (19.298)
  Month 26 - SF36 VT (Sweden): number analyzed (Participants) | 1652
  Month 26 - SF36 VT (Sweden) | 71.78 (20.945)
  Month 26 - SF36 SF (Sweden): number analyzed (Participants) | 1653
  Month 26 - SF36 SF (Sweden) | 90.58 (18.238)
  Month 26 - SF36 RE (Sweden): number analyzed (Participants) | 1655
  Month 26 - SF36 RE (Sweden) | 90.08 (18.878)
  Month 26 - SF36 MH (Sweden): number analyzed (Participants) | 1652
  Month 26 - SF36 MH (Sweden) | 85.22 (15.521)
  Month 38 - SF36 PF (Sweden): number analyzed (Participants) | 1628
  Month 38 - SF36 PF (Sweden) | 79.20 (21.873)
  Month 38 - SF36 RP (Sweden): number analyzed (Participants) | 1626
  Month 38 - SF36 RP (Sweden) | 82.09 (25.357)
  Month 38 - SF36 BP (Sweden): number analyzed (Participants) | 1626
  Month 38 - SF36 BP (Sweden) | 74.38 (24.731)
  Month 38 - SF36 GH (Sweden): number analyzed (Participants) | 1630
  Month 38 - SF36 GH (Sweden) | 74.19 (19.653)
  Month 38 - SF36 VT (Sweden): number analyzed (Participants) | 1627
  Month 38 - SF36 VT (Sweden) | 70.77 (21.471)
  Month 38 - SF36 SF (Sweden): number analyzed (Participants) | 1627
  Month 38 - SF36 SF (Sweden) | 90.26 (18.614)
  Month 38 - SF36 RE (Sweden): number analyzed (Participants) | 1626
  Month 38 - SF36 RE (Sweden) | 88.83 (20.313)
  Month 38 - SF36 MH (Sweden): number analyzed (Participants) | 1627
  Month 38 - SF36 MH (Sweden) | 84.81 (15.910)
  Month 0 - SF36 PF (Taiwan): number analyzed (Participants) | 2382
  Month 0 - SF36 PF (Taiwan) | 83.07 (20.550)
  Month 0 - SF36 RP (Taiwan): number analyzed (Participants) | 2382
  Month 0 - SF36 RP (Taiwan) | 83.88 (21.920)
  Month 0 - SF36 BP (Taiwan): number analyzed (Participants) | 2381
  Month 0 - SF36 BP (Taiwan) | 83.37 (19.421)
  Month 0 - SF36 GH (Taiwan): number analyzed (Participants) | 2382
  Month 0 - SF36 GH (Taiwan) | 70.15 (18.885)
  Month 0 - SF36 VT (Taiwan): number analyzed (Participants) | 2380
  Month 0 - SF36 VT (Taiwan) | 72.29 (18.430)
  Month 0 - SF36 SF (Taiwan): number analyzed (Participants) | 2381
  Month 0 - SF36 SF (Taiwan) | 90.41 (14.557)
  Month 0 - SF36 RE (Taiwan): number analyzed (Participants) | 2382
  Month 0 - SF36 RE (Taiwan) | 86.56 (19.473)
  Month 0 - SF36 MH (Taiwan): number analyzed (Participants) | 2380
  Month 0 - SF36 MH (Taiwan) | 78.06 (16.593)
  Month 14 - SF36 PF (Taiwan): number analyzed (Participants) | 2246
  Month 14 - SF36 PF (Taiwan) | 83.38 (18.693)
  Month 14 - SF36 RP (Taiwan): number analyzed (Participants) | 2246
  Month 14 - SF36 RP (Taiwan) | 82.95 (22.339)
  Month 14 - SF36 BP (Taiwan): number analyzed (Participants) | 2246
  Month 14 - SF36 BP (Taiwan) | 81.58 (20.215)
  Month 14 - SF36 GH (Taiwan): number analyzed (Participants) | 2246
  Month 14 - SF36 GH (Taiwan) | 69.11 (19.118)
  Month 14 - SF36 VT (Taiwan): number analyzed (Participants) | 2246
  Month 14 - SF36 VT (Taiwan) | 70.03 (19.270)
  Month 14 - SF36 SF (Taiwan): number analyzed (Participants) | 2246
  Month 14 - SF36 SF (Taiwan) | 89.74 (15.538)
  Month 14 - SF36 RE (Taiwan): number analyzed (Participants) | 2246
  Month 14 - SF36 RE (Taiwan) | 84.98 (19.686)
  Month 14 - SF36 MH (Taiwan): number analyzed (Participants) | 2246
  Month 14 - SF36 MH (Taiwan) | 77.42 (16.610)
  Month 26 - SF36 PF (Taiwan): number analyzed (Participants) | 2188
  Month 26 - SF36 PF (Taiwan) | 82.08 (19.937)
  Month 26 - SF36 RP (Taiwan): number analyzed (Participants) | 2188
  Month 26 - SF36 RP (Taiwan) | 82.18 (23.207)
  Month 26 - SF36 BP (Taiwan): number analyzed (Participants) | 2187
  Month 26 - SF36 BP (Taiwan) | 80.84 (20.720)
  Month 26 - SF36 GH (Taiwan): number analyzed (Participants) | 2188
  Month 26 - SF36 GH (Taiwan) | 68.56 (20.296)
  Month 26 - SF36 VT (Taiwan): number analyzed (Participants) | 2187
  Month 26 - SF36 VT (Taiwan) | 70.04 (19.068)
  Month 26 - SF36 SF (Taiwan): number analyzed (Participants) | 2187
  Month 26 - SF36 SF (Taiwan) | 89.70 (15.829)
  Month 26 - SF36 RE (Taiwan): number analyzed (Participants) | 2188
  Month 26 - SF36 RE (Taiwan) | 84.86 (20.402)
  Month 26 - SF36 MH (Taiwan): number analyzed (Participants) | 2187
  Month 26 - SF36 MH (Taiwan) | 77.00 (17.208)
  Month 38 - SF36 PF (Taiwan): number analyzed (Participants) | 2104
  Month 38 - SF36 PF (Taiwan) | 80.62 (21.330)
  Month 38 - SF36 RP (Taiwan): number analyzed (Participants) | 2105
  Month 38 - SF36 RP (Taiwan) | 78.40 (25.194)
  Month 38 - SF36 BP (Taiwan): number analyzed (Participants) | 2105
  Month 38 - SF36 BP (Taiwan) | 79.55 (21.425)
  Month 38 - SF36 GH (Taiwan): number analyzed (Participants) | 2106
  Month 38 - SF36 GH (Taiwan) | 67.12 (20.107)
  Month 38 - SF36 VT (Taiwan): number analyzed (Participants) | 2104
  Month 38 - SF36 VT (Taiwan) | 68.57 (19.453)
  Month 38 - SF36 SF (Taiwan): number analyzed (Participants) | 2105
  Month 38 - SF36 SF (Taiwan) | 87.10 (17.663)
  Month 38 - SF36 RE (Taiwan): number analyzed (Participants) | 2105
  Month 38 - SF36 RE (Taiwan) | 81.25 (22.276)
  Month 38 - SF36 MH (Taiwan): number analyzed (Participants) | 2104
  Month 38 - SF36 MH (Taiwan) | 76.20 (17.290)
  Month 0 - SF36 PF (United Kingdom): number analyzed (Participants) | 1293
  Month 0 - SF36 PF (United Kingdom) | 71.71 (27.696)
  Month 0 - SF36 RP (United Kingdom): number analyzed (Participants) | 1294
  Month 0 - SF36 RP (United Kingdom) | 79.47 (26.123)
  Month 0 - SF36 BP (United Kingdom): number analyzed (Participants) | 1301
  Month 0 - SF36 BP (United Kingdom) | 73.04 (26.098)
  Month 0 - SF36 GH (United Kingdom): number analyzed (Participants) | 1303
  Month 0 - SF36 GH (United Kingdom) | 71.43 (19.664)
  Month 0 - SF36 VT (United Kingdom): number analyzed (Participants) | 1301
  Month 0 - SF36 VT (United Kingdom) | 64.93 (20.355)
  Month 0 - SF36 SF (United Kingdom): number analyzed (Participants) | 1303
  Month 0 - SF36 SF (United Kingdom) | 88.02 (21.772)
  Month 0 - SF36 RE (United Kingdom): number analyzed (Participants) | 1293
  Month 0 - SF36 RE (United Kingdom) | 87.82 (22.674)
  Month 0 - SF36 MH (United Kingdom): number analyzed (Participants) | 1301
  Month 0 - SF36 MH (United Kingdom) | 80.46 (17.348)
  Month 14 - SF36 PF (United Kingdom): number analyzed (Participants) | 1228
  Month 14 - SF36 PF (United Kingdom) | 68.78 (29.011)
  Month 14 - SF36 RP (United Kingdom): number analyzed (Participants) | 1229
  Month 14 - SF36 RP (United Kingdom) | 73.59 (30.401)
  Month 14 - SF36 BP (United Kingdom): number analyzed (Participants) | 1233
  Month 14 - SF36 BP (United Kingdom) | 68.88 (27.303)
  Month 14 - SF36 GH (United Kingdom): number analyzed (Participants) | 1238
  Month 14 - SF36 GH (United Kingdom) | 67.55 (21.359)
  Month 14 - SF36 VT (United Kingdom): number analyzed (Participants) | 1234
  Month 14 - SF36 VT (United Kingdom) | 60.94 (21.934)
  Month 14 - SF36 SF (United Kingdom): number analyzed (Participants) | 1234
  Month 14 - SF36 SF (United Kingdom) | 85.18 (24.093)
  Month 14 - SF36 RE (United Kingdom): number analyzed (Participants) | 1227
  Month 14 - SF36 RE (United Kingdom) | 85.24 (25.645)
  Month 14 - SF36 MH (United Kingdom): number analyzed (Participants) | 1233
  Month 14 - SF36 MH (United Kingdom) | 79.24 (18.331)
  Month 26 - SF36 PF (United Kingdom): number analyzed (Participants) | 1179
  Month 26 - SF36 PF (United Kingdom) | 67.69 (28.942)
  Month 26 - SF36 RP (United Kingdom): number analyzed (Participants) | 1179
  Month 26 - SF36 RP (United Kingdom) | 72.59 (29.682)
  Month 26 - SF36 BP (United Kingdom): number analyzed (Participants) | 1188
  Month 26 - SF36 BP (United Kingdom) | 67.81 (27.447)
  Month 26 - SF36 GH (United Kingdom): number analyzed (Participants) | 1189
  Month 26 - SF36 GH (United Kingdom) | 67.53 (21.378)
  Month 26 - SF36 VT (United Kingdom): number analyzed (Participants) | 1189
  Month 26 - SF36 VT (United Kingdom) | 59.99 (22.567)
  Month 26 - SF36 SF (United Kingdom): number analyzed (Participants) | 1189
  Month 26 - SF36 SF (United Kingdom) | 82.92 (26.021)
  Month 26 - SF36 RE (United Kingdom): number analyzed (Participants) | 1178
  Month 26 - SF36 RE (United Kingdom) | 83.17 (26.731)
  Month 26 - SF36 MH (United Kingdom): number analyzed (Participants) | 1189
  Month 26 - SF36 MH (United Kingdom) | 78.18 (19.361)
  Month 38 - SF36 PF (United Kingdom): number analyzed (Participants) | 1162
  Month 38 - SF36 PF (United Kingdom) | 66.64 (28.795)
  Month 38 - SF36 RP (United Kingdom): number analyzed (Participants) | 1162
  Month 38 - SF36 RP (United Kingdom) | 71.46 (29.715)
  Month 38 - SF36 BP (United Kingdom): number analyzed (Participants) | 1162
  Month 38 - SF36 BP (United Kingdom) | 67.74 (27.445)
  Month 38 - SF36 GH (United Kingdom): number analyzed (Participants) | 1166
  Month 38 - SF36 GH (United Kingdom) | 67.39 (20.666)
  Month 38 - SF36 VT (United Kingdom): number analyzed (Participants) | 1165
  Month 38 - SF36 VT (United Kingdom) | 59.64 (21.532)
  Month 38 - SF36 SF (United Kingdom): number analyzed (Participants) | 1165
  Month 38 - SF36 SF (United Kingdom) | 82.92 (24.958)
  Month 38 - SF36 RE (United Kingdom): number analyzed (Participants) | 1162
  Month 38 - SF36 RE (United Kingdom) | 83.37 (25.844)
  Month 38 - SF36 MH (United Kingdom): number analyzed (Participants) | 1165
  Month 38 - SF36 MH (United Kingdom) | 78.61 (18.453)
  Month 0 - SF36 PF (United States): number analyzed (Participants) | 3114
  Month 0 - SF36 PF (United States) | 76.45 (23.632)
  Month 0 - SF36 RP (United States): number analyzed (Participants) | 3132
  Month 0 - SF36 RP (United States) | 81.58 (23.473)
  Month 0 - SF36 BP (United States): number analyzed (Participants) | 3118
  Month 0 - SF36 BP (United States) | 75.20 (21.417)
  Month 0 - SF36 GH (United States): number analyzed (Participants) | 3139
  Month 0 - SF36 GH (United States) | 78.06 (16.471)
  Month 0 - SF36 VT (United States): number analyzed (Participants) | 3138
  Month 0 - SF36 VT (United States) | 69.99 (17.564)
  Month 0 - SF36 SF (United States): number analyzed (Participants) | 3120
  Month 0 - SF36 SF (United States) | 92.28 (16.120)
  Month 0 - SF36 RE (United States): number analyzed (Participants) | 3133
  Month 0 - SF36 RE (United States) | 90.44 (18.574)
  Month 0 - SF36 MH (United States): number analyzed (Participants) | 3138
  Month 0 - SF36 MH (United States) | 84.73 (13.554)
  Month 14 - SF36 PF (United States): number analyzed (Participants) | 2812
  Month 14 - SF36 PF (United States) | 74.70 (25.252)
  Month 14 - SF36 RP (United States): number analyzed (Participants) | 2825
  Month 14 - SF36 RP (United States) | 78.58 (26.202)
  Month 14 - SF36 BP (United States): number analyzed (Participants) | 2804
  Month 14 - SF36 BP (United States) | 73.02 (23.499)
  Month 14 - SF36 GH (United States): number analyzed (Participants) | 2829
  Month 14 - SF36 GH (United States) | 75.44 (17.797)
  Month 14 - SF36 VT (United States): number analyzed (Participants) | 2817
  Month 14 - SF36 VT (United States) | 67.13 (18.980)
  Month 14 - SF36 SF (United States): number analyzed (Participants) | 2813
  Month 14 - SF36 SF (United States) | 89.99 (18.818)
  Month 14 - SF36 RE (United States): number analyzed (Participants) | 2825
  Month 14 - SF36 RE (United States) | 88.06 (21.433)
  Month 14 - SF36 MH (United States): number analyzed (Participants) | 2817
  Month 14 - SF36 MH (United States) | 83.61 (14.733)
  Month 26 - SF36 PF (United States): number analyzed (Participants) | 2669
  Month 26 - SF36 PF (United States) | 73.93 (25.438)
  Month 26 - SF36 RP (United States): number analyzed (Participants) | 2682
  Month 26 - SF36 RP (United States) | 78.00 (26.125)
  Month 26 - SF36 BP (United States): number analyzed (Participants) | 2650
  Month 26 - SF36 BP (United States) | 73.01 (23.580)
  Month 26 - SF36 GH (United States): number analyzed (Participants) | 2685
  Month 26 - SF36 GH (United States) | 74.92 (18.181)
  Month 26 - SF36 VT (United States): number analyzed (Participants) | 2658
  Month 26 - SF36 VT (United States) | 66.95 (19.411)
  Month 26 - SF36 SF (United States): number analyzed (Participants) | 2674
  Month 26 - SF36 SF (United States) | 89.94 (19.038)
  Month 26 - SF36 RE (United States): number analyzed (Participants) | 2681
  Month 26 - SF36 RE (United States) | 87.83 (21.258)
  Month 26 - SF36 MH (United States): number analyzed (Participants) | 2658
  Month 26 - SF36 MH (United States) | 83.48 (15.118)
  Month 38 - SF36 PF (United States): number analyzed (Participants) | 2518
  Month 38 - SF36 PF (United States) | 71.66 (26.334)
  Month 38 - SF36 RP (United States): number analyzed (Participants) | 2526
  Month 38 - SF36 RP (United States) | 75.97 (26.785)
  Month 38 - SF36 BP (United States): number analyzed (Participants) | 2518
  Month 38 - SF36 BP (United States) | 71.31 (23.682)
  Month 38 - SF36 GH (United States): number analyzed (Participants) | 2530
  Month 38 - SF36 GH (United States) | 73.23 (18.699)
  Month 38 - SF36 VT (United States): number analyzed (Participants) | 2526
  Month 38 - SF36 VT (United States) | 65.74 (19.480)
  Month 38 - SF36 SF (United States): number analyzed (Participants) | 2526
  Month 38 - SF36 SF (United States) | 88.78 (19.795)
  Month 38 - SF36 RE (United States): number analyzed (Participants) | 2526
  Month 38 - SF36 RE (United States) | 87.28 (22.058)
  Month 38 - SF36 MH (United States): number analyzed (Participants) | 2526
  Month 38 - SF36 MH (United States) | 83.20 (15.151)

2. Secondary Outcome: Distribution of EuroQol (EQ)-5D Questionnaire Scale Scores, by Country
Description: The EQ-5D questionnaire is a generic measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D defines health in terms of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each item has 3 possible responses (No symptoms, Moderate symptoms, Extreme symptoms). The 5 items are then combined to generate health profiles that are subsequently converted to a continuous single index utility score using a one to one matching. Country or region-specific value sets are used for the score conversion. The scores range from less than 0 (where 0 is the value of a health state equivalent to dead) to 1 (the value of full health), with higher scores indicating higher health utility.
  The EQ-5D also contains a visual analogue scale (VAS). The VAS records the respondent's self-rated health on a vertical scale, ranging from 0(worst imaginable health state) to 100(best imaginable health state).
Time Frame: At Month 0, 14, 26 and 38
Population: Analysis was performed on all subjects included in the Total Vaccinated Cohort (TVC) of Zoster-064
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Overall Group
Number analyzed (Participants) | 3128
Scale score
  Month 0 - EQ5D Utility (Australia): number analyzed (Participants) | 479
  Month 0 - EQ5D Utility (Australia) | 0.8072 (0.19966)
  Month 0 - EQ5D VAS (Australia): number analyzed (Participants) | 478
  Month 0 - EQ5D VAS (Australia) | 85.43 (13.031)
  Month 14 - EQ5D Utility (Australia): number analyzed (Participants) | 431
  Month 14 - EQ5D Utility (Australia) | 0.7671 (0.19586)
  Month 14 - EQ5D VAS (Australia): number analyzed (Participants) | 424
  Month 14 - EQ5D VAS (Australia) | 81.48 (14.544)
  Month 26 - EQ5D Utility (Australia): number analyzed (Participants) | 412
  Month 26 - EQ5D Utility (Australia) | 0.7582 (0.20781)
  Month 26 - EQ5D VAS (Australia): number analyzed (Participants) | 410
  Month 26 - EQ5D VAS (Australia) | 81.24 (16.066)
  Month 38 - EQ5D Utility (Australia): number analyzed (Participants) | 402
  Month 38 - EQ5D Utility (Australia) | 0.7589 (0.19839)
  Month 38 - EQ5D VAS (Australia): number analyzed (Participants) | 401
  Month 38 - EQ5D VAS (Australia) | 80.86 (15.135)
  Month 0 - EQ5D Utility (Brazil): number analyzed (Participants) | 1239
  Month 0 - EQ5D Utility (Brazil) | 0.8565 (0.14387)
  Month 0 - EQ5D VAS (Brazil): number analyzed (Participants) | 1249
  Month 0 - EQ5D VAS (Brazil) | 82.92 (15.561)
  Month 14 - EQ5D Utility (Brazil): number analyzed (Participants) | 1146
  Month 14 - EQ5D Utility (Brazil) | 0.8524 (0.14637)
  Month 14 - EQ5D VAS (Brazil): number analyzed (Participants) | 1145
  Month 14 - EQ5D VAS (Brazil) | 81.57 (16.303)
  Month 26 - EQ5D Utility (Brazil): number analyzed (Participants) | 1115
  Month 26 - EQ5D Utility (Brazil) | 0.8535 (0.14893)
  Month 26 - EQ5D VAS (Brazil): number analyzed (Participants) | 1117
  Month 26 - EQ5D VAS (Brazil) | 81.96 (15.919)
  Month 38 - EQ5D Utility (Brazil): number analyzed (Participants) | 1094
  Month 38 - EQ5D Utility (Brazil) | 0.8410 (0.16028)
  Month 38 - EQ5D VAS (Brazil): number analyzed (Participants) | 1094
  Month 38 - EQ5D VAS (Brazil) | 81.41 (16.253)
  Month 0 - EQ5D Utility (Canada): number analyzed (Participants) | 1379
  Month 0 - EQ5D Utility (Canada) | 0.8894 (0.12153)
  Month 0 - EQ5D VAS (Canada): number analyzed (Participants) | 1383
  Month 0 - EQ5D VAS (Canada) | 83.75 (12.586)
  Month 14 - EQ5D Utility (Canada): number analyzed (Participants) | 1335
  Month 14 - EQ5D Utility (Canada) | 0.8647 (0.14416)
  Month 14 - EQ5D VAS (Canada): number analyzed (Participants) | 1339
  Month 14 - EQ5D VAS (Canada) | 81.59 (13.743)
  Month 26 - EQ5D Utility (Canada): number analyzed (Participants) | 1283
  Month 26 - EQ5D Utility (Canada) | 0.8649 (0.13286)
  Month 26 - EQ5D VAS (Canada): number analyzed (Participants) | 1287
  Month 26 - EQ5D VAS (Canada) | 81.03 (14.370)
  Month 38 - EQ5D Utility (Canada): number analyzed (Participants) | 1247
  Month 38 - EQ5D Utility (Canada) | 0.8515 (0.13904)
  Month 38 - EQ5D VAS (Canada): number analyzed (Participants) | 1251
  Month 38 - EQ5D VAS (Canada) | 80.23 (15.018)
  Month 0 - EQ5D Utility (Czechia): number analyzed (Participants) | 1226
  Month 0 - EQ5D Utility (Czechia) | 0.8724 (0.13090)
  Month 0 - EQ5D VAS (Czechia): number analyzed (Participants) | 1226
  Month 0 - EQ5D VAS (Czechia) | 83.60 (13.604)
  Month 14 - EQ5D Utility (Czechia): number analyzed (Participants) | 1210
  Month 14 - EQ5D Utility (Czechia) | 0.8214 (0.16054)
  Month 14 - EQ5D VAS (Czechia): number analyzed (Participants) | 1210
  Month 14 - EQ5D VAS (Czechia) | 83.61 (15.134)
  Month 26 - EQ5D Utility (Czechia): number analyzed (Participants) | 1199
  Month 26 - EQ5D Utility (Czechia) | 0.8034 (0.16000)
  Month 26 - EQ5D VAS (Czechia): number analyzed (Participants) | 1199
  Month 26 - EQ5D VAS (Czechia) | 81.24 (15.485)
  Month 38 - EQ5D Utility (Czechia): number analyzed (Participants) | 1177
  Month 38 - EQ5D Utility (Czechia) | 0.8080 (0.16581)
  Month 38 - EQ5D VAS (Czechia): number analyzed (Participants) | 1177
  Month 38 - EQ5D VAS (Czechia) | 81.88 (15.349)
  Month 0 - EQ5D Utility (Estonia): number analyzed (Participants) | 2120
  Month 0 - EQ5D Utility (Estonia) | 0.8393 (0.13827)
  Month 0 - EQ5D VAS (Estonia): number analyzed (Participants) | 2121
  Month 0 - EQ5D VAS (Estonia) | 71.57 (16.882)
  Month 14 - EQ5D Utility (Estonia): number analyzed (Participants) | 2056
  Month 14 - EQ5D Utility (Estonia) | 0.7796 (0.16461)
  Month 14 - EQ5D VAS (Estonia): number analyzed (Participants) | 2058
  Month 14 - EQ5D VAS (Estonia) | 71.61 (17.646)
  Month 26 - EQ5D Utility (Estonia): number analyzed (Participants) | 2025
  Month 26 - EQ5D Utility (Estonia) | 0.7176 (0.17669)
  Month 26 - EQ5D VAS (Estonia): number analyzed (Participants) | 2030
  Month 26 - EQ5D VAS (Estonia) | 66.39 (19.086)
  Month 38 - EQ5D Utility (Estonia): number analyzed (Participants) | 1991
  Month 38 - EQ5D Utility (Estonia) | 0.6800 (0.16682)
  Month 38 - EQ5D VAS (Estonia): number analyzed (Participants) | 1992
  Month 38 - EQ5D VAS (Estonia) | 64.89 (18.325)
  Month 0 - EQ5D Utility (Finland): number analyzed (Participants) | 2993
  Month 0 - EQ5D Utility (Finland) | 0.8767 (0.15909)
  Month 0 - EQ5D VAS (Finland): number analyzed (Participants) | 2977
  Month 0 - EQ5D VAS (Finland) | 83.57 (11.773)
  Month 14 - EQ5D Utility (Finland): number analyzed (Participants) | 2893
  Month 14 - EQ5D Utility (Finland) | 0.8415 (0.17068)
  Month 14 - EQ5D VAS (Finland): number analyzed (Participants) | 2918
  Month 14 - EQ5D VAS (Finland) | 81.15 (13.553)
  Month 26 - EQ5D Utility (Finland): number analyzed (Participants) | 2828
  Month 26 - EQ5D Utility (Finland) | 0.8367 (0.17273)
  Month 26 - EQ5D VAS (Finland): number analyzed (Participants) | 2846
  Month 26 - EQ5D VAS (Finland) | 80.89 (13.565)
  Month 38 - EQ5D Utility (Finland): number analyzed (Participants) | 2794
  Month 38 - EQ5D Utility (Finland) | 0.8249 (0.17615)
  Month 38 - EQ5D VAS (Finland): number analyzed (Participants) | 2807
  Month 38 - EQ5D VAS (Finland) | 80.22 (13.795)
  Month 0 - EQ5D Utility (France): number analyzed (Participants) | 1086
  Month 0 - EQ5D Utility (France) | 0.8266 (0.20137)
  Month 0 - EQ5D VAS (France): number analyzed (Participants) | 1088
  Month 0 - EQ5D VAS (France) | 74.39 (15.885)
  Month 14 - EQ5D Utility (France): number analyzed (Participants) | 1060
  Month 14 - EQ5D Utility (France) | 0.8139 (0.22983)
  Month 14 - EQ5D VAS (France): number analyzed (Participants) | 1055
  Month 14 - EQ5D VAS (France) | 73.30 (15.614)
  Month 26 - EQ5D Utility (France): number analyzed (Participants) | 986
  Month 26 - EQ5D Utility (France) | 0.8094 (0.23680)
  Month 26 - EQ5D VAS (France): number analyzed (Participants) | 975
  Month 26 - EQ5D VAS (France) | 72.97 (16.001)
  Month 38 - EQ5D Utility (France): number analyzed (Participants) | 977
  Month 38 - EQ5D Utility (France) | 0.7981 (0.24427)
  Month 38 - EQ5D VAS (France): number analyzed (Participants) | 977
  Month 38 - EQ5D VAS (France) | 73.44 (15.264)
  Month 0 - EQ5D Utility (Germany): number analyzed (Participants) | 1910
  Month 0 - EQ5D Utility (Germany) | 0.8877 (0.16705)
  Month 0 - EQ5D VAS (Germany): number analyzed (Participants) | 1905
  Month 0 - EQ5D VAS (Germany) | 77.11 (17.322)
  Month 14 - EQ5D Utility (Germany): number analyzed (Participants) | 1793
  Month 14 - EQ5D Utility (Germany) | 0.8644 (0.18635)
  Month 14 - EQ5D VAS (Germany): number analyzed (Participants) | 1803
  Month 14 - EQ5D VAS (Germany) | 74.09 (18.406)
  Month 26 - EQ5D Utility (Germany): number analyzed (Participants) | 1759
  Month 26 - EQ5D Utility (Germany) | 0.8561 (0.19313)
  Month 26 - EQ5D VAS (Germany): number analyzed (Participants) | 1764
  Month 26 - EQ5D VAS (Germany) | 72.47 (18.917)
  Month 38 - EQ5D Utility (Germany): number analyzed (Participants) | 1692
  Month 38 - EQ5D Utility (Germany) | 0.8335 (0.20997)
  Month 38 - EQ5D VAS (Germany): number analyzed (Participants) | 1697
  Month 38 - EQ5D VAS (Germany) | 70.79 (19.049)
  Month 0 - EQ5D Utility (Hong Kong): number analyzed (Participants) | 648
  Month 0 - EQ5D Utility (Hong Kong) | 0.8743 (0.14053)
  Month 0 - EQ5D VAS (Hong Kong): number analyzed (Participants) | 648
  Month 0 - EQ5D VAS (Hong Kong) | 82.32 (12.502)
  Month 14 - EQ5D Utility (Hong Kong): number analyzed (Participants) | 620
  Month 14 - EQ5D Utility (Hong Kong) | 0.8398 (0.15518)
  Month 14 - EQ5D VAS (Hong Kong): number analyzed (Participants) | 622
  Month 14 - EQ5D VAS (Hong Kong) | 81.14 (13.191)
  Month 26 - EQ5D Utility (Hong Kong): number analyzed (Participants) | 601
  Month 26 - EQ5D Utility (Hong Kong) | 0.8463 (0.15796)
  Month 26 - EQ5D VAS (Hong Kong): number analyzed (Participants) | 604
  Month 26 - EQ5D VAS (Hong Kong) | 79.65 (14.173)
  Month 38 - EQ5D Utility (Hong Kong): number analyzed (Participants) | 595
  Month 38 - EQ5D Utility (Hong Kong) | 0.8393 (0.15566)
  Month 38 - EQ5D VAS (Hong Kong): number analyzed (Participants) | 595
  Month 38 - EQ5D VAS (Hong Kong) | 80.61 (13.669)
  Month 0 - EQ5D Utility (Italy): number analyzed (Participants) | 276
  Month 0 - EQ5D Utility (Italy) | 0.8219 (0.14860)
  Month 0 - EQ5D VAS (Italy): number analyzed (Participants) | 275
  Month 0 - EQ5D VAS (Italy) | 79.80 (13.270)
  Month 14 - EQ5D Utility (Italy): number analyzed (Participants) | 261
  Month 14 - EQ5D Utility (Italy) | 0.8383 (0.13899)
  Month 14 - EQ5D VAS (Italy): number analyzed (Participants) | 260
  Month 14 - EQ5D VAS (Italy) | 79.72 (13.041)
  Month 26 - EQ5D Utility (Italy): number analyzed (Participants) | 250
  Month 26 - EQ5D Utility (Italy) | 0.8398 (0.14228)
  Month 26 - EQ5D VAS (Italy): number analyzed (Participants) | 251
  Month 26 - EQ5D VAS (Italy) | 78.84 (12.701)
  Month 38 - EQ5D Utility (Italy): number analyzed (Participants) | 242
  Month 38 - EQ5D Utility (Italy) | 0.8173 (0.16055)
  Month 38 - EQ5D VAS (Italy): number analyzed (Participants) | 241
  Month 38 - EQ5D VAS (Italy) | 77.19 (14.648)
  Month 0 - EQ5D Utility (Japan): number analyzed (Participants) | 770
  Month 0 - EQ5D Utility (Japan) | 0.9139 (0.13118)
  Month 0 - EQ5D VAS (Japan): number analyzed (Participants) | 771
  Month 0 - EQ5D VAS (Japan) | 80.43 (12.559)
  Month 14 - EQ5D Utility (Japan): number analyzed (Participants) | 737
  Month 14 - EQ5D Utility (Japan) | 0.9011 (0.13948)
  Month 14 - EQ5D VAS (Japan): number analyzed (Participants) | 738
  Month 14 - EQ5D VAS (Japan) | 81.53 (12.924)
  Month 26 - EQ5D Utility (Japan): number analyzed (Participants) | 721
  Month 26 - EQ5D Utility (Japan) | 0.8899 (0.13631)
  Month 26 - EQ5D VAS (Japan): number analyzed (Participants) | 723
  Month 26 - EQ5D VAS (Japan) | 81.76 (13.591)
  Month 38 - EQ5D Utility (Japan): number analyzed (Participants) | 702
  Month 38 - EQ5D Utility (Japan) | 0.8946 (0.14504)
  Month 38 - EQ5D VAS (Japan): number analyzed (Participants) | 702
  Month 38 - EQ5D VAS (Japan) | 80.65 (13.332)
  Month 0 - EQ5D Utility (Republic of Korea): number analyzed (Participants) | 1063
  Month 0 - EQ5D Utility (Republic of Korea) | 0.8263 (0.16773)
  Month 0 - EQ5D VAS (Republic of Korea): number analyzed (Participants) | 1064
  Month 0 - EQ5D VAS (Republic of Korea) | 79.81 (13.754)
  Month 14 - EQ5D Utility (Republic of Korea): number analyzed (Participants) | 939
  Month 14 - EQ5D Utility (Republic of Korea) | 0.8050 (0.17430)
  Month 14 - EQ5D VAS (Republic of Korea): number analyzed (Participants) | 940
  Month 14 - EQ5D VAS (Republic of Korea) | 76.95 (15.411)
  Month 26 - EQ5D Utility (Republic of Korea): number analyzed (Participants) | 904
  Month 26 - EQ5D Utility (Republic of Korea) | 0.8120 (0.16588)
  Month 26 - EQ5D VAS (Republic of Korea): number analyzed (Participants) | 904
  Month 26 - EQ5D VAS (Republic of Korea) | 76.53 (14.551)
  Month 38 - EQ5D Utility (Republic of Korea): number analyzed (Participants) | 860
  Month 38 - EQ5D Utility (Republic of Korea) | 0.8140 (0.18373)
  Month 38 - EQ5D VAS (Republic of Korea): number analyzed (Participants) | 858
  Month 38 - EQ5D VAS (Republic of Korea) | 75.97 (14.418)
  Month 0 - EQ5D Utility (Mexico): number analyzed (Participants) | 926
  Month 0 - EQ5D Utility (Mexico) | 0.8863 (0.13315)
  Month 0 - EQ5D VAS (Mexico): number analyzed (Participants) | 924
  Month 0 - EQ5D VAS (Mexico) | 83.57 (13.337)
  Month 14 - EQ5D Utility (Mexico): number analyzed (Participants) | 818
  Month 14 - EQ5D Utility (Mexico) | 0.8733 (0.14923)
  Month 14 - EQ5D VAS (Mexico): number analyzed (Participants) | 812
  Month 14 - EQ5D VAS (Mexico) | 83.11 (13.943)
  Month 26 - EQ5D Utility (Mexico): number analyzed (Participants) | 783
  Month 26 - EQ5D Utility (Mexico) | 0.8615 (0.16050)
  Month 26 - EQ5D VAS (Mexico): number analyzed (Participants) | 773
  Month 26 - EQ5D VAS (Mexico) | 81.96 (16.173)
  Month 38 - EQ5D Utility (Mexico): number analyzed (Participants) | 747
  Month 38 - EQ5D Utility (Mexico) | 0.8465 (0.16123)
  Month 38 - EQ5D VAS (Mexico): number analyzed (Participants) | 745
  Month 38 - EQ5D VAS (Mexico) | 80.49 (17.163)
  Month 0 - EQ5D Utility (Spain): number analyzed (Participants) | 1977
  Month 0 - EQ5D Utility (Spain) | 0.8827 (0.19725)
  Month 0 - EQ5D VAS (Spain): number analyzed (Participants) | 1986
  Month 0 - EQ5D VAS (Spain) | 79.44 (16.744)
  Month 14 - EQ5D Utility (Spain): number analyzed (Participants) | 1838
  Month 14 - EQ5D Utility (Spain) | 0.8372 (0.23163)
  Month 14 - EQ5D VAS (Spain): number analyzed (Participants) | 1846
  Month 14 - EQ5D VAS (Spain) | 75.42 (17.281)
  Month 26 - EQ5D Utility (Spain): number analyzed (Participants) | 1784
  Month 26 - EQ5D Utility (Spain) | 0.8265 (0.24231)
  Month 26 - EQ5D VAS (Spain): number analyzed (Participants) | 1792
  Month 26 - EQ5D VAS (Spain) | 75.71 (16.869)
  Month 38 - EQ5D Utility (Spain): number analyzed (Participants) | 1736
  Month 38 - EQ5D Utility (Spain) | 0.8236 (0.24430)
  Month 38 - EQ5D VAS (Spain): number analyzed (Participants) | 1743
  Month 38 - EQ5D VAS (Spain) | 74.97 (17.471)
  Month 0 - EQ5D Utility (Sweden): number analyzed (Participants) | 1733
  Month 0 - EQ5D Utility (Sweden) | 0.8527 (0.13410)
  Month 0 - EQ5D VAS (Sweden): number analyzed (Participants) | 1726
  Month 0 - EQ5D VAS (Sweden) | 85.05 (12.622)
  Month 14 - EQ5D Utility (Sweden): number analyzed (Participants) | 1667
  Month 14 - EQ5D Utility (Sweden) | 0.8387 (0.14270)
  Month 14 - EQ5D VAS (Sweden): number analyzed (Participants) | 1671
  Month 14 - EQ5D VAS (Sweden) | 82.31 (14.782)
  Month 26 - EQ5D Utility (Sweden): number analyzed (Participants) | 1644
  Month 26 - EQ5D Utility (Sweden) | 0.8371 (0.14325)
  Month 26 - EQ5D VAS (Sweden): number analyzed (Participants) | 1641
  Month 26 - EQ5D VAS (Sweden) | 82.19 (14.924)
  Month 38 - EQ5D Utility (Sweden): number analyzed (Participants) | 1619
  Month 38 - EQ5D Utility (Sweden) | 0.8191 (0.14856)
  Month 38 - EQ5D VAS (Sweden): number analyzed (Participants) | 1618
  Month 38 - EQ5D VAS (Sweden) | 81.11 (15.993)
  Month 0 - EQ5D Utility (Taiwan): number analyzed (Participants) | 2377
  Month 0 - EQ5D Utility (Taiwan) | 0.9159 (0.12941)
  Month 0 - EQ5D VAS (Taiwan): number analyzed (Participants) | 2380
  Month 0 - EQ5D VAS (Taiwan) | 83.20 (11.888)
  Month 14 - EQ5D Utility (Taiwan): number analyzed (Participants) | 2241
  Month 14 - EQ5D Utility (Taiwan) | 0.9114 (0.13530)
  Month 14 - EQ5D VAS (Taiwan): number analyzed (Participants) | 2245
  Month 14 - EQ5D VAS (Taiwan) | 82.25 (12.466)
  Month 26 - EQ5D Utility (Taiwan): number analyzed (Participants) | 2179
  Month 26 - EQ5D Utility (Taiwan) | 0.9018 (0.14211)
  Month 26 - EQ5D VAS (Taiwan): number analyzed (Participants) | 2187
  Month 26 - EQ5D VAS (Taiwan) | 82.88 (12.412)
  Month 38 - EQ5D Utility (Taiwan): number analyzed (Participants) | 2095
  Month 38 - EQ5D Utility (Taiwan) | 0.8927 (0.15029)
  Month 38 - EQ5D VAS (Taiwan): number analyzed (Participants) | 2100
  Month 38 - EQ5D VAS (Taiwan) | 81.61 (12.684)
  Month 0 - EQ5D Utility (United Kingdom): number analyzed (Participants) | 1291
  Month 0 - EQ5D Utility (United Kingdom) | 0.8069 (0.22841)
  Month 0 - EQ5D VAS (United Kingdom): number analyzed (Participants) | 1296
  Month 0 - EQ5D VAS (United Kingdom) | 79.37 (16.162)
  Month 14 - EQ5D Utility (United Kingdom): number analyzed (Participants) | 1225
  Month 14 - EQ5D Utility (United Kingdom) | 0.7743 (0.26018)
  Month 14 - EQ5D VAS (United Kingdom): number analyzed (Participants) | 1227
  Month 14 - EQ5D VAS (United Kingdom) | 77.47 (17.954)
  Month 26 - EQ5D Utility (United Kingdom): number analyzed (Participants) | 1179
  Month 26 - EQ5D Utility (United Kingdom) | 0.7535 (0.27379)
  Month 26 - EQ5D VAS (United Kingdom): number analyzed (Participants) | 1180
  Month 26 - EQ5D VAS (United Kingdom) | 76.58 (18.074)
  Month 38 - EQ5D Utility (United Kingdom): number analyzed (Participants) | 1162
  Month 38 - EQ5D Utility (United Kingdom) | 0.7569 (0.26046)
  Month 38 - EQ5D VAS (United Kingdom): number analyzed (Participants) | 1163
  Month 38 - EQ5D VAS (United Kingdom) | 76.98 (17.609)
  Month 0 - EQ5D Utility (United States): number analyzed (Participants) | 3112
  Month 0 - EQ5D Utility (United States) | 0.8843 (0.12499)
  Month 0 - EQ5D VAS (United States) | 85.22 (12.555)
  Month 14 - EQ5D Utility (United States): number analyzed (Participants) | 2795
  Month 14 - EQ5D Utility (United States) | 0.8747 (0.14000)
  Month 14 - EQ5D VAS (United States): number analyzed (Participants) | 2799
  Month 14 - EQ5D VAS (United States) | 84.06 (14.054)
  Month 26 - EQ5D Utility (United States): number analyzed (Participants) | 2644
  Month 26 - EQ5D Utility (United States) | 0.8722 (0.13899)
  Month 26 - EQ5D VAS (United States): number analyzed (Participants) | 2659
  Month 26 - EQ5D VAS (United States) | 83.63 (14.344)
  Month 38 - EQ5D Utility (United States): number analyzed (Participants) | 2507
  Month 38 - EQ5D Utility (United States) | 0.8576 (0.14879)
  Month 38 - EQ5D VAS (United States): number analyzed (Participants) | 2514
  Month 38 - EQ5D VAS (United States) | 82.75 (14.788)

3. Primary Outcome: Number of Subjects by Frailty Status, at Baseline
Description: Frailty status was measured in relation to the accumulation of deficits using a Frailty Index (FI) adapted from the model proposed by Mitnitski et al. [Mitnitski, 2001]. The different aspects of frailty composing the FI were assessed through the medical history and components of the Short Form 36 Questionnaire (SF-36) and EuroQol (EQ)-5D questionnaires recorded pre-vaccination Dose 1 (in the study ZOSTER-006[NCT01165177] and ZOSTER-022[NCT01165229]).
  If the FI was less than or equal to 0.08, the subject was classified as Non-Frail. If the score was greater than 0.08 but less than or equal to 0.25, the subject was classified as pre-frail. If the score was greater than 0.25, the subject was classified as Frail. Subjects without a FI score were classified as unknown.
Time Frame: At Baseline (Month 0)
Population: Analysis was performed on all subjects included in the Total Vaccinated Cohort (TVC) of Zoster-064
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Group
Number analyzed (Participants) | 26976
Participants
  Non-Frail | 11518
  Pre-Frail | 12290
  Frail | 3037
  Unknown | 131

4. Secondary Outcome: Incidence Rate (Per 1000 Person-years) of Confirmed Herpes Zoster (HZ) Cases, by Frailty Status
Description: Incidence rate (IR) of confirmed Herpes zoster (HZ) cases with 95% Confidence Interval (CI) calculated as the number of cases per 1000 person-years : numerator = number of confirmed HZ cases reported during the follow-up (FU) period at risk; denominator = total Person-years at risk, i.e. sum of FU periods at risk expressed in years until first confirmed HZ cases or occurrence of treatment for relapse. A suspected HZ case defined as (1) new rash characteristic of HZ (e.g., unilateral, dermatomal and accompanied by pain broadly defined to include allodynia, pruritus or other sensations), or vesicular rash suggestive of Varicella Zoster Virus (VZV) infection regardless of the distribution, and no alternative diagnosis; or (2) clinical presentation and specific laboratory findings suggestive of VZV infection in the absence of HZ or VZV rash. A suspected case of HZ was confirmed either by PCR or by the HZ Ascertainment Committee (HZAC), consisting of physicians with HZ expertise.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: Analysis was performed on all subjects in the Modified Total Vaccinated Cohort (mTVC) of ZOSTER-064. The Z-064 mTVC excluded subjects in the Z-064 TVC who were not administered the second vaccination or who developed a confirmed case of Herpes Zoster (HZ) prior to 1 month after the second vaccination.
Measure: Number; unit: Cases per 1000 person-year
Groups:
- Non-Frail-HZ/su: Adults aged ≥50 years of age who received HZ/su vaccine (in Zoster-006/022 study) and were categorized as non-frail.
- Non-Frail-Placebo: Adults aged ≥50 years of age who received placebo (in Zoster-006/022 study) and were categorized as non-frail.
- Pre-Frail-HZ/su: Adults aged ≥50 years of age who received HZ/su vaccine (in Zoster-006/022 study) and were categorized as pre-frail.
- Pre-Frail-Placebo: Adults aged ≥50 years of age who received placebo (in Zoster-006/022 study) and were categorized as pre-frail.
- Frail-HZ/su: Adults aged ≥50 years of age who received HZ/su vaccine (in Zoster-006/022 study) and were categorized as frail.
- Frail-Placebo: Adults aged ≥50 years of age who received placebo (in Zoster-006/022 study) and were categorized as frail.
- Unknown-HZ/su: Adults aged ≥50 years of age who received HZ/su vaccine (in Zoster-006/022 study) and were not assigned a frailty category.
- Unknown-Placebo: Adults aged ≥50 years of age who received placebo (in Zoster-006/022 study) and were not assigned a frailty category.
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
Number analyzed (Participants) | 5545 | 5551 | 5738 | 5969 | 1449 | 1348 | 53 | 62
Cases per 1000 person-year | 0.4 | 8.8 | 0.8 | 8.6 | 1.0 | 9.9 | 0.0 | 25.8
Statistical Analysis 1: Comparison: Non-Frail-HZ/su vs Non-Frail-Placebo; Efficacy analysis aimed at comparing the confimed herpes zoster for Herpes Zoster incidence rate between Non-Frail-HZ/su vs Non-Frail-Placebo groups; Test type: Other — Vaccine efficacy rate was calculated as 100*(1-RR) with RR=relative risk of developing the confimed herpes zoster for Herpes Zoster subunit vaccine Group compared to Placebo Group; p < 0.0001, Poisson exact test; Vaccine Efficacy rate = 95.81, 95% CI 2-sided [91.58 to 98.22]
Statistical Analysis 2: Comparison: Pre-Frail-HZ/su vs Pre-Frail-Placebo; Efficacy analysis aimed at comparing the confimed herpes zoster for Herpes Zoster incidence rate between Pre-Frail-HZ/su vs Pre-Frail-Placebo groups; Test type: Other — Vaccine efficacy rate was calculated as 100*(1-RR) with RR=relative risk of developing the confimed herpes zoster for Herpes Zoster subunit vaccine group compared to placebo people; p < 0.0001, Poisson exact test; Vaccine Efficacy rate = 90.4, 95% CI 2-sided [84.41 to 94.43]
Statistical Analysis 3: Comparison: Frail-HZ/su vs Frail-Placebo; Efficacy analysis aimed at comparing the confimed herpes zoster for Herpes Zoster incidence rate between Frail-HZ/su vs Frail-Placebo groups; Test type: Other — [test comment as in outcome 4, analysis 2]; p < 0.0001, Poisson exact test; Vaccine Efficacy rate = 90.17, 95% CI 2-sided [75.36 to 96.65]
Statistical Analysis 4: Comparison: Unknown-HZ/su vs Unknown-Placebo; Efficacy analysis aimed at comparing the confimed herpes zoster for Herpes Zoster incidence rate between Unknown-HZ/su vs Unknown-Placebo groups; Test type: Other — [test comment as in outcome 4, analysis 2]; p = 0.069, Poisson exact test; Vaccine Efficacy rate = 100, 95% CI 2-sided [14.61 to 100]

5. Secondary Outcome: Herpes Zoster Burden of Illness Score, by Frailty Status
Description: Zoster Brief Pain Inventory (ZBPI) Burden of Illness (BOI) score was calculated as the sum of the ZBPI worst pain scores for all subjects in the group divided by the total follow-up time (Person-years). HZ Burden of Illness score for subjects was calculated from the Zoster Brief Pain Inventory (ZBPI), for each confirmed HZ cases responding to the "worst pain" question in both ZOSTER-006 and ZOSTER-022, and defined as the area under the curve of confirmed HZ-associated pain plotted against time during the 182-day period after the onset of the case. Subjects who developed HZ presented "burden-of-illness" scores ranging from 0 up to, theoretically, 1820. A score of 0 is recorded for subjects in whom HZ did not develop during the study period. Subjects who had a confirmed Zoster episode but who did not have at least 1 ZBPI assessment were excluded from the analysis.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 4
Measure: Number; unit: Score per subject-year
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
Number analyzed (Participants) | 5545 | 5550 | 5738 | 5968 | 1449 | 1348 | 53 | 60
Score per subject-year | 0.017 | 1.173 | 0.108 | 1.475 | 0.345 | 2.330 | 0.000 | 3.303
Statistical Analysis 1: Comparison: Non-Frail-HZ/su vs Non-Frail-Placebo; VE against confirmed HZ BOI and 95% confidence intervals (CIs) are presented by frailty status in the mTVC; Test type: Other — VE against the BOI due to HZ (VE BOI ) was defined as the relative reduction in the BOI score in the vaccine group as compared with that in the placebo group and calculated as 1 - relative risk (i.e., 1- the HZ BOI score in the vaccine group divided by the HZ BOI score in the placebo group); Vaccine Efficacy rate = 98.6, 95% CI 2-sided [97.1 to 100]
Statistical Analysis 2: Comparison: Pre-Frail-HZ/su vs Pre-Frail-Placebo; VE against confirmed HZ BOI and 95% confidence intervals (CIs) are presented by frailty status in the mTVC; Test type: Other — [test comment as in outcome 5, analysis 1]; Vaccine Efficacy rate = 92.6, 95% CI 2-sided [86.6 to 98.7]
Statistical Analysis 3: Comparison: Frail-HZ/su vs Frail-Placebo; VE against confirmed HZ BOI and 95% confidence intervals (CIs) are presented by frailty status in the mTVC; Test type: Other — [test comment as in outcome 5, analysis 1]; Vaccine Efficacy rate = 85.2, 95% CI 2-sided [62.6 to 100]
Statistical Analysis 4: Comparison: Unknown-HZ/su vs Unknown-Placebo; VE against the BOI due to confirmed HZ. The 95% Confidence Interval was not calculated as there were no subjects reported with a confirmed Zoster episode in the Unknown-HZ/su Group; Test type: Other — [test comment as in outcome 5, analysis 1]; Vaccine Efficacy rate = 100

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms, by Frailty Status
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within 7 days (Days 0-6) after each vaccination
Population: Analysis was performed on all subjects in the Zoster-064 TVC diary card subset for analysis of reactogenicity. Note that due to the retrospective observational nature of this study, new safety data was not collected in Zoster-064; the safety data presented here was originally collected as part of the Zoster-006 and Zoster-022 studies.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
Number analyzed (Participants) | 2007 | 2034 | 1977 | 1964 | 489 | 468 | 21 | 17
Participants
  Any Pain | 1655 | 209 | 1494 | 211 | 322 | 51 | 17 | 1
  Grade 3 Pain | 115 | 4 | 125 | 6 | 38 | 5 | 1 | 0
  Any Redness | 805 | 25 | 734 | 28 | 160 | 2 | 11 | 0
  Grade 3 Redness | 75 | 0 | 46 | 0 | 12 | 0 | 0 | 0
  Any Swelling | 545 | 18 | 497 | 22 | 107 | 3 | 6 | 1
  Grade 3 Swelling | 24 | 0 | 19 | 0 | 2 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms, by Frailty Status
Description: Assessed solicited general symptoms were, fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], headache, myalgia, shivering and gastro-intestinal (GI) symptoms(nausea, vomiting, diarrhoea and/or abdominal pain) Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within 7 days (Days 0-6) after each vaccination
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
Number analyzed (Participants) | 2007 | 2034 | 1971 | 1964 | 488 | 468 | 21 | 18
Participants
  Any Fatigue | 951 | 301 | 848 | 339 | 164 | 96 | 5 | 4
  Grade 3 Fatigue | 114 | 15 | 93 | 17 | 22 | 8 | 0 | 0
  Related Fatigue | 848 | 233 | 715 | 231 | 139 | 54 | 5 | 4
  Any Gastrointestinal symptoms | 369 | 157 | 325 | 166 | 65 | 56 | 2 | 2
  Grade 3 Gastrointestinal symptoms | 26 | 11 | 28 | 8 | 6 | 5 | 0 | 0
  Related Gastrointestinal symptoms | 298 | 88 | 229 | 86 | 44 | 26 | 0 | 2
  Any Headache | 838 | 287 | 676 | 311 | 147 | 89 | 6 | 3
  Grade 3 Headache | 74 | 8 | 53 | 12 | 17 | 10 | 0 | 0
  Related Headache | 735 | 202 | 582 | 198 | 122 | 59 | 5 | 3
  Any Myalgia | 952 | 209 | 828 | 225 | 173 | 75 | 5 | 2
  Grade 3 Myalgia | 100 | 8 | 89 | 8 | 28 | 12 | 0 | 0
  Related Myalgia | 864 | 153 | 730 | 172 | 148 | 47 | 4 | 2
  Any Shivering | 623 | 111 | 459 | 107 | 86 | 41 | 3 | 3
  Grade 3 Shivering | 103 | 4 | 57 | 6 | 18 | 2 | 0 | 0
  Related Shivering | 559 | 80 | 398 | 74 | 74 | 22 | 3 | 3
  Any Fever | 465 | 52 | 368 | 55 | 70 | 19 | 1 | 0
  Grade 3 Fever | 6 | 4 | 5 | 3 | 2 | 0 | 0 | 0
  Related Fever | 419 | 35 | 316 | 29 | 57 | 8 | 1 | 0

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs), by Frailty Status
Description: An unsolicited AE covered any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 30 days (Days 0 - 29) after each vaccination
Population: Analysis was performed on all subjects included in the Zoster-064 TVC. Note that due to the retrospective observational nature of this study, new safety data was not collected in Zoster-064; the safety data presented here was originally collected as part of the Zoster-006 and Zoster-022 studies.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
Number analyzed (Participants) | 5784 | 5734 | 6071 | 6219 | 1573 | 1464 | 59 | 72
Participants
  Any AE | 2984 | 1696 | 3019 | 2034 | 754 | 520 | 23 | 22
  Grade 3 AE | 429 | 182 | 429 | 242 | 134 | 80 | 5 | 5
  Related AE | 2223 | 386 | 1962 | 420 | 449 | 91 | 16 | 6

9. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs), by Frailty Status
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Related SAEs were those considered vaccine-related by the investigator.
Time Frame: From Month 0 to Month 14
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
Number analyzed (Participants) | 5784 | 5734 | 6071 | 6219 | 1573 | 1464 | 59 | 72
Participants
  Any SAEs | 357 | 328 | 697 | 751 | 293 | 332 | 8 | 10
  Related SAEs | 6 | 3 | 6 | 9 | 2 | 0 | 0 | 0

10. Secondary Outcome: Number of Subjects With SAEs Related to Study Participation or to a Concurrent GSK Medication/Vaccine, by Frailty Status
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Related SAEs throughout the entire study period by frailty status were reported for SAEs considered related to study participation or to a concurrent GSK medication/vaccine.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
Number analyzed (Participants) | 5784 | 5734 | 6071 | 6219 | 1573 | 1464 | 59 | 72
Participants | 14 | 16 | 55 | 49 | 24 | 31 | 0 | 2

11. Secondary Outcome: Number of Subjects With Any Fatal Serious Adverse Events (SAEs), by Frailty Status
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
Number analyzed (Participants) | 5784 | 5734 | 6071 | 6219 | 1573 | 1464 | 59 | 72
Participants | 124 | 109 | 299 | 343 | 174 | 182 | 2 | 6

12. Secondary Outcome: Number of Subjects With Any and Related Potential Immune-mediated Diseases (pIMDs), by Frailty Status
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Related = pIMDs assessed by the investigator as related to the vaccination.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
Number analyzed (Participants) | 5784 | 5734 | 6071 | 6219 | 1573 | 1464 | 59 | 72
Participants
  Any pIMDs | 74 | 69 | 76 | 90 | 15 | 27 | 1 | 0
  Related pIMDs | 4 | 7 | 9 | 6 | 2 | 1 | 0 | 0

13. Secondary Outcome: Anti-glycoprotein E (Anti-gE) Antibody (Ab) Concentrations, by Frailty Status, in a Subset of Subjects
Description: Anti-gE Ab concentrations as determined by Enzyme-linked Immunosorbent Assay (ELISA), in a subset of subjects. The assay cut-off is 97 milli-international units (mIU)/mL.
Time Frame: Pre-vaccination at Month 0, and post second dose at Months 3, 14, 26 and 38
Population: Analysis was performed on a subset of subjects in Z-064 According to Protocol (ATP) cohort for immunogenicity-humoral (i.e. those among the Z-064 TVC, who met all eligibility criteria, complied with procedures and intervals for analysis,with no elimination criteria during Z-006/022 studies,and for whom data concerning immunogenicity were available)
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
Number analyzed (Participants) | 603 | 606 | 655 | 697 | 138 | 125 | 4 | 4
mIU/mL
  Anti-gE Ab at Month 0: number analyzed (Participants) | 603 | 606 | 653 | 695 | 138 | 125 | 4 | 4
  Anti-gE Ab at Month 0 | 1251.6 [1151.7 to 1360.3] | 1389.1 [1286.6 to 1499.8] | 1363.0 [1262.1 to 1471.9] | 1325.4 [1227.0 to 1431.7] | 1450.8 [1230.9 to 1710.1] | 1457.7 [1213.6 to 1750.8] | 1172.9 [389.0 to 3536.5] | 836.2 [157.6 to 4434.9]
  Anti-gE antibody at Month 3 | 53120.8 [50229.2 to 56178.8] | 1314.6 [1211.8 to 1426.2] | 52514.0 [49937.0 to 55224.0] | 1266.9 [1171.6 to 1369.9] | 44914.9 [39734.6 to 50770.6] | 1310.8 [1089.8 to 1576.7] | 34703.5 [18272.8 to 65908.6] | 854.8 [119.2 to 6132.2]
  Anti-gE antibody at Month 14: number analyzed (Participants) | 591 | 586 | 640 | 662 | 124 | 114 | 4 | 4
  Anti-gE antibody at Month 14 | 18628.2 [17477.6 to 19854.6] | 1272.4 [1174.4 to 1378.5] | 16689.7 [15739.5 to 17697.2] | 1224.7 [1129.9 to 1327.4] | 13405.4 [11701.3 to 15357.7] | 1337.8 [1089.7 to 1642.4] | 9834.3 [3469.9 to 27871.7] | 888.2 [270.6 to 2914.9]
  Anti-gE antibody at Month 26: number analyzed (Participants) | 582 | 571 | 617 | 628 | 115 | 112 | 4 | 3
  Anti-gE antibody at Month 26 | 14502.0 [13610.9 to 15451.4] | 1355.5 [1253.2 to 1466.1] | 13344.2 [12592.6 to 14140.6] | 1320.2 [1219.1 to 1429.6] | 11060.6 [9689.0 to 12626.3] | 1431.4 [1156.2 to 1772.2] | 5278.7 [1248.8 to 22313.6] | 712.8 [143.6 to 3538.1]
  Anti-gE antibody at Month 38: number analyzed (Participants) | 555 | 553 | 586 | 588 | 110 | 109 | 4 | 3
  Anti-gE antibody at Month 38 | 12505.4 [11695.1 to 13371.8] | 1304.3 [1203.5 to 1413.5] | 11099.9 [10458.8 to 11780.4] | 1274.3 [1171.4 to 1386.2] | 8694.8 [7612.1 to 9931.6] | 1399.1 [1112.6 to 1759.2] | 5128.7 [1349.3 to 19494.2] | 614.9 [64.5 to 5863.9]

14. Secondary Outcome: Anti-Varicella Zoster Virus (Anti-VZV) Antibody (Ab) Concentrations, by Frailty Status, in a Subset of Subjects
Description: Anti-VZV Ab concentrations as determined by Enzyme-linked Immunosorbent Assay (ELISA), in a subset of subjects. The assay cut-off is 25 mIU/mL.
Time Frame: Pre-vaccination at Month 0, and post second dose at Months 3, 14, 26 and 38
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
Number analyzed (Participants) | 603 | 594 | 655 | 677 | 138 | 124 | 4 | 4
mIU/mL
  Anti-VZV antibody at Month 0: number analyzed (Participants) | 588 | 587 | 643 | 676 | 135 | 124 | 4 | 4
  Anti-VZV antibody at Month 0 | 966.9 [893.6 to 1046.2] | 1053.3 [981.8 to 1130.0] | 992.9 [927.8 to 1062.7] | 1036.9 [969.7 to 1108.7] | 996.6 [866.7 to 1146.1] | 1054.7 [894.9 to 1243.1] | 712.3 [166.2 to 3052.9] | 553.7 [63.7 to 4812.0]
  Anti-VZV antibody at Month 3: number analyzed (Participants) | 603 | 594 | 655 | 677 | 138 | 121 | 4 | 4
  Anti-VZV antibody at Month 3 | 9206.0 [8731.3 to 9706.5] | 989.8 [922.5 to 1061.9] | 9468.9 [9046.7 to 9910.8] | 997.0 [933.4 to 1065.0] | 8162.4 [7332.5 to 9086.2] | 904.2 [764.4 to 1069.4] | 6499.1 [4054.7 to 10417.1] | 601.7 [78.7 to 4601.0]
  Anti-VZV antibody at Month 14: number analyzed (Participants) | 587 | 579 | 636 | 649 | 124 | 114 | 4 | 4
  Anti-VZV antibody at Month 14 | 3791.4 [3569.3 to 4027.2] | 931.4 [867.4 to 1000.1] | 3630.9 [3450.2 to 3821.0] | 945.3 [883.8 to 1011.0] | 3034.4 [2719.3 to 3386.1] | 921.9 [769.0 to 1105.2] | 2175.3 [1073.6 to 4407.6] | 646.9 [90.1 to 4646.3]
  Anti-VZV antibody at Month 26: number analyzed (Participants) | 580 | 554 | 615 | 610 | 115 | 112 | 4 | 3
  Anti-VZV antibody at Month 26 | 3226.8 [3037.6 to 3427.7] | 986.0 [918.0 to 1058.9] | 3261.7 [3094.9 to 3437.5] | 1040.8 [973.8 to 1112.3] | 2759.4 [2472.4 to 3079.8] | 1023.0 [850.1 to 1231.1] | 1909.4 [839.1 to 4344.8] | 374.7 [48.9 to 2869.2]
  Anti-VZV antibody at Month 38: number analyzed (Participants) | 550 | 526 | 578 | 575 | 109 | 109 | 4 | 3
  Anti-VZV antibody at Month 38 | 3111.6 [2928.2 to 3306.4] | 1029.2 [958.8 to 1104.8] | 2966.3 [2813.9 to 3126.9] | 1068.0 [994.7 to 1146.7] | 2462.1 [2201.7 to 2753.4] | 1098.1 [903.3 to 1334.8] | 1928.4 [857.8 to 4335.2] | 286.3 [33.3 to 2460.0]

ADVERSE EVENTS:
Time Frame: Solicited symptoms: within 7 days (Days 0-6) after vaccination; Unsolicited adverse events: within 30 days (Days 0-29) after vaccination; Serious Adverse Events (SAEs): during the entire study period (3 to 5 year period following Day 0).
Description: Note that due to the retrospective observational nature of this study, new safety data was not collected in Zoster-064; the safety data presented here was originally collected as part of the Zoster-006 and Zoster-022 studies.
Arm/Group | Non-Frail-HZ/su | Non-Frail-Placebo | Pre-Frail-HZ/su | Pre-Frail-Placebo | Frail-HZ/su | Frail-Placebo | Unknown-HZ/su | Unknown-Placebo
All-Cause Mortality (participants affected / at risk) | 124/5784 | 109/5734 | 299/6071 | 343/6219 | 174/1573 | 182/1464 | 2/59 | 6/72
Serious Adverse Events (participants affected / at risk) | 453/5784 | 413/5734 | 886/6071 | 964/6219 | 385/1573 | 426/1464 | 10/59 | 14/72
Other Adverse Events (participants affected / at risk) | 2961/5784 | 1668/5734 | 2955/6071 | 1953/6219 | 730/1573 | 481/1464 | 23/59 | 22/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Frail-HZ/su (N=5784) | Non-Frail-Placebo (N=5734) | Pre-Frail-HZ/su (N=6071) | Pre-Frail-Placebo (N=6219) | Frail-HZ/su (N=1573) | Frail-Placebo (N=1464) | Unknown-HZ/su (N=59) | Unknown-Placebo (N=72)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 6 (6) | 9 (9) | 3 (3) | 5 (7) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (3) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia vitamin b12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pernicious anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0) | 4 (4) | 5 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 6 (6) | 15 (16) | 24 (24) | 7 (7) | 16 (17) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (3) | 0 (0) | 5 (5) | 2 (2) | 7 (7) | 6 (6) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 3 (3) | 1 (1) | 4 (4) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2) | 7 (7) | 4 (4) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 12 (12) | 12 (12) | 28 (36) | 33 (33) | 16 (17) | 10 (12) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0) | 5 (5) | 2 (2) | 2 (2) | 6 (6) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 5 (5) | 1 (1) | 15 (15) | 16 (16) | 8 (8) | 7 (7) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 9 (9) | 4 (4) | 37 (37) | 43 (46) | 23 (25) | 30 (35) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 3 (3) | 11 (11) | 14 (16) | 17 (17) | 21 (23) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular deconditioning (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 6 (6) | 8 (8) | 17 (18) | 20 (20) | 14 (14) | 13 (15) | 1 (1) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 8 (8) | 17 (17) | 35 (35) | 33 (33) | 18 (19) | 19 (19) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 4 (5) | 1 (1) | 7 (7) | 20 (20) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 3 (3) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy alcoholic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronotropic incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystic fibrosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 3 (3) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 2 (2) | 7 (7) | 7 (7) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Macular cyst (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 4 (4) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (6) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 7 (7) | 4 (4) | 7 (7) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (5) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (5) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 7 (9) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal cyst (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 6 (6) | 2 (2) | 16 (16) | 20 (20) | 5 (5) | 3 (6) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 5 (5) | 8 (8) | 14 (14) | 20 (20) | 8 (8) | 14 (14) | 0 (0) | 1 (1)
Drowning (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 1 (1) | 9 (9) | 4 (4) | 3 (3) | 7 (7) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Strangulated hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 4 (4) | 2 (2) | 8 (8) | 5 (5) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis in device (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Choroidal effusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iridocele (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lens dislocation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular vascular disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis alcoholic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 5 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gingival disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal congestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mesenteric artery embolism (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic artery aneurysm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device deposit issue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gravitational oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyp (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device battery issue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device leakage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 4 (4) | 7 (8) | 12 (14) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 1 (1) | 5 (5) | 5 (5) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 8 (8) | 6 (6) | 8 (8) | 13 (13) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatty liver alcoholic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder perforation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic granulomatous angiitis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyloidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 4 (4) | 5 (5) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 5 (5) | 3 (4) | 4 (4) | 8 (8) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 5 (5) | 3 (3) | 7 (7) | 8 (8) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 9 (10) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 5 (5) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2) | 6 (7) | 7 (7) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis caliciviral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal gangrene (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroborreliosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 20 (20) | 17 (17) | 55 (57) | 50 (52) | 27 (29) | 32 (36) | 2 (2) | 2 (2)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purulence (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 1 (1) | 4 (4) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 4 (4) | 8 (9) | 14 (14) | 16 (16) | 10 (11) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 6 (6) | 4 (4) | 7 (7) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Serratia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shigella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tularaemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 4 (4) | 18 (19) | 20 (21) | 11 (14) | 8 (10) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 2 (2) | 4 (5) | 5 (5) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visceral leishmaniasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcaligenes infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerotic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cavernous sinus thrombosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis a (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Incision site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 6 (6) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psittacosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic shock syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fistula infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candiduria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Graft infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mycobacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory moniliasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 6 (6) | 4 (4) | 4 (4) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrical burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 5 (5) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0) | 5 (5) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 6 (6) | 14 (14) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 4 (4) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Kidney contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) | 8 (8) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 6 (6) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (4) | 5 (5) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood heavy metal increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye penetration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve root injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aneurysm perforation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 7 (7) | 2 (2) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (6) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (6) | 7 (7) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Marasmus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5) | 14 (14) | 14 (14) | 10 (10) | 7 (7) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (5) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Still's disease adult onset (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Adult t-cell lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4) | 3 (3) | 13 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 3 (3) | 2 (2) | 6 (6) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 7 (7) | 5 (5) | 7 (7) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 7 (7) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 4 (4) | 16 (16) | 11 (11) | 7 (8) | 4 (4) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 3 (3) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 7 (7) | 5 (5) | 8 (9) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 12 (12) | 16 (16) | 10 (10) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaplastic thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioimmunoblastic t-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse large b-cell lymphoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant fibrous histiocytoma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant lymphoma unclassifiable high grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant mast cell neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of ampulla of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Metastases to gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basilar artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 5 (5) | 9 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 8 (8) | 2 (2) | 14 (14) | 16 (17) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 7 (7) | 11 (11) | 27 (27) | 21 (22) | 16 (16) | 8 (9) | 1 (1) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 6 (6) | 4 (4) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuritis cranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 4 (4) | 9 (9) | 13 (14) | 2 (2) | 9 (10) | 0 (0) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 3 (3) | 17 (18) | 9 (9) | 6 (7) | 7 (9) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viiith nerve lesion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain stem syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral artery thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drop attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dural arteriovenous fistula (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspraxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miller fisher syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mixed dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mononeuritis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post polio syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Senile dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia with lewy bodies (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Progressive supranuclear palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal claudication (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Korsakoff's syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Schizoaffective disorder bipolar type (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somatoform disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breathing-related sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium febrile (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 2 (2) | 14 (14) | 11 (11) | 6 (7) | 10 (11) | 0 (0) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (5) | 2 (2) | 11 (11) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 5 (5) | 6 (6) | 6 (6) | 5 (6) | 0 (0) | 0 (0)
Renal hypertension (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral polyp (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis interstitial (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephroangiosclerosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal artery occlusion (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 (5) | 3 (3) | 4 (4) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine enlargement (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 6 (8) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 10 (11) | 8 (8) | 15 (20) | 15 (17) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (4) | 8 (8) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 12 (12) | 22 (22) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 10 (10) | 12 (12) | 10 (10) | 5 (5) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural calcification (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary bulla (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aneurysm ruptured (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic rupture (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (4) | 3 (3) | 6 (6) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 5 (5) | 16 (16) | 16 (18) | 5 (5) | 14 (15) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 3 (3) | 1 (1) | 2 (2) | 7 (7) | 4 (5) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Internal haemorrhage (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyarteritis nodosa (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporal arteritis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angiodysplasia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic dilatation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Inferior vena caval occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Microscopic polyangiitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose ulceration (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Labile hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboangiitis obliterans (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Frail-HZ/su (N=5784) | Non-Frail-Placebo (N=5734) | Pre-Frail-HZ/su (N=6071) | Pre-Frail-Placebo (N=6219) | Frail-HZ/su (N=1573) | Frail-Placebo (N=1464) | Unknown-HZ/su (N=59) | Unknown-Placebo (N=72)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 6 (6) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 9 (10) | 2 (2) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (3) | 2 (2) | 6 (6) | 9 (9) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 6 (7) | 5 (5) | 11 (11) | 6 (6) | 3 (3) | 1 (1) | 1 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malformation venous (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 15 (15) | 7 (8) | 6 (8) | 6 (7) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Eustachian tube disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 4 (4) | 4 (4) | 7 (7) | 7 (7) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 14 (15) | 7 (8) | 22 (22) | 21 (23) | 6 (7) | 8 (9) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Androgen deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basedow's disease (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypogonadism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 3 (3) | 2 (2) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 2 (3) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 3 (3) | 6 (6) | 6 (6) | 13 (13) | 6 (6) | 5 (5) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chorioretinal atrophy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chorioretinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromatopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 4 (4) | 4 (4) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 4 (4) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dark circles under eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 4 (4) | 2 (2) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enophthalmos (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 4 (4) | 4 (4) | 8 (8) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid rash (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelids pruritus (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation decreased (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Narrow anterior chamber angle (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 4 (4) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic vein thrombosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panophthalmitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal degeneration (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy hypertensive (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichiasis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 4 (4) | 5 (6) | 8 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 3 (3) | 7 (7) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 17 (18) | 12 (14) | 15 (15) | 13 (13) | 4 (4) | 6 (7) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 23 (25) | 28 (30) | 23 (24) | 32 (34) | 6 (6) | 5 (5) | 1 (2) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acid peptic disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aerophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aptyalism (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 3 (4) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (10) | 12 (13) | 18 (18) | 13 (14) | 6 (6) | 7 (7) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 56 (59) | 41 (43) | 50 (52) | 53 (55) | 18 (18) | 13 (14) | 1 (1) | 1 (2)
Diverticulum (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 1 (1) | 8 (8) | 10 (10) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 14 (15) | 11 (11) | 15 (18) | 16 (18) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (2) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 9 (11) | 6 (8) | 15 (17) | 11 (11) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 5 (6) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 8 (8) | 10 (10) | 9 (9) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 9 (9) | 11 (11) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanosis coli (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 7 (7) | 5 (5) | 7 (8) | 5 (5) | 3 (3) | 4 (4) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 92 (104) | 28 (36) | 71 (80) | 32 (34) | 18 (21) | 8 (8) | 0 (0) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oesophageal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 5 (6) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatic steatosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary gland cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue blistering (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth deposit (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth erosion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 22 (23) | 25 (25) | 13 (13) | 21 (22) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 26 (27) | 10 (10) | 18 (18) | 17 (20) | 9 (9) | 7 (7) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Administration site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 38 (41) | 6 (6) | 26 (28) | 13 (13) | 8 (9) | 3 (3) | 0 (0) | 2 (2)
Axillary pain (General disorders) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 3 (3) | 2 (2) | 6 (6) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 10 (11) | 10 (12) | 19 (20) | 9 (10) | 3 (5) | 5 (6) | 0 (0) | 0 (0)
Chills (General disorders) | 252 (297) | 16 (17) | 189 (218) | 14 (15) | 36 (41) | 2 (2) | 3 (4) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device breakage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 3 (4) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 252 (300) | 47 (49) | 182 (216) | 75 (78) | 34 (44) | 8 (8) | 2 (2) | 1 (2)
Feeling abnormal (General disorders) | 5 (6) | 2 (2) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 28 (30) | 4 (4) | 20 (22) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 27 (30) | 2 (2) | 16 (16) | 7 (7) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Implant site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 61 (78) | 21 (21) | 39 (43) | 18 (20) | 8 (10) | 3 (3) | 0 (0) | 0 (0)
Injection site atrophy (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 16 (19) | 16 (17) | 16 (16) | 13 (15) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Injection site coldness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 10 (10) | 2 (2) | 9 (9) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Injection site eczema (General disorders) | 3 (4) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 607 (819) | 14 (14) | 535 (700) | 22 (24) | 115 (139) | 1 (2) | 4 (4) | 0 (0)
Injection site haematoma (General disorders) | 9 (9) | 5 (7) | 4 (4) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 5 (5) | 6 (6) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site hyperaesthesia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site hypersensitivity (General disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site hypoaesthesia (General disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 21 (23) | 2 (2) | 25 (29) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 19 (21) | 0 (0) | 21 (22) | 1 (1) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Injection site injury (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site irritation (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site joint pain (General disorders) | 21 (25) | 1 (1) | 22 (22) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site lymphadenopathy (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site macule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 3 (3) | 1 (1) | 5 (6) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site movement impairment (General disorders) | 4 (4) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 12 (14) | 0 (0) | 20 (21) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1454 (2157) | 94 (110) | 1334 (1877) | 109 (119) | 298 (404) | 29 (34) | 8 (12) | 3 (3)
Injection site papule (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site paraesthesia (General disorders) | 2 (2) | 3 (3) | 2 (3) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 144 (170) | 11 (13) | 115 (140) | 16 (17) | 36 (39) | 3 (3) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 30 (32) | 1 (1) | 22 (24) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 27 (31) | 4 (4) | 27 (31) | 7 (7) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 455 (587) | 8 (8) | 390 (490) | 8 (8) | 88 (112) | 4 (6) | 2 (2) | 0 (0)
Injection site ulcer (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site vesicles (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 63 (68) | 0 (0) | 66 (75) | 4 (4) | 12 (14) | 0 (0) | 1 (2) | 0 (0)
Injury associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 5 (5) | 7 (8) | 2 (2) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 113 (126) | 19 (20) | 87 (99) | 16 (16) | 20 (21) | 3 (3) | 1 (1) | 1 (1)
Metaplasia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucous membrane disorder (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 1 (1) | 5 (5) | 6 (6) | 3 (3) | 7 (7) | 1 (1) | 0 (0)
Pain (General disorders) | 98 (114) | 10 (10) | 71 (76) | 17 (18) | 17 (19) | 4 (4) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 4 (4) | 3 (3) | 6 (6) | 5 (5) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Polyp (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 560 (678) | 33 (35) | 341 (410) | 29 (30) | 58 (67) | 5 (5) | 2 (3) | 0 (0)
Reactogenicity event (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sluggishness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcer haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site coldness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site discolouration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 12 (16) | 0 (0) | 19 (23) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Vaccination site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site inflammation (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 30 (37) | 0 (0) | 25 (29) | 5 (5) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Vaccination site pruritus (General disorders) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site reaction (General disorders) | 5 (7) | 0 (0) | 8 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site swelling (General disorders) | 8 (11) | 0 (0) | 9 (9) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Vaccination site warmth (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to chemicals (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to plants (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 6 (7) | 9 (9) | 7 (8) | 7 (7) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (3) | 1 (1) | 4 (6) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute tonsillitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alveolar osteitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blastocystis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Borrelia infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 24 (24) | 32 (32) | 60 (63) | 41 (41) | 16 (17) | 15 (15) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 5 (5) | 10 (10) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic hepatitis b (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 7 (7) | 4 (4) | 11 (11) | 19 (20) | 11 (11) | 8 (8) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 14 (14) | 10 (11) | 17 (18) | 15 (16) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatophytosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 3 (3) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 6 (6) | 7 (7) | 6 (6) | 5 (5) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema migrans (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 18 (19) | 20 (20) | 19 (19) | 15 (15) | 1 (1) | 7 (7) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 7 (7) | 5 (5) | 9 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 5 (5) | 7 (7) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
H1n1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoid infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 15 (18) | 20 (21) | 9 (10) | 7 (8) | 7 (7) | 4 (4) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected bites (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected varicose vein (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 30 (31) | 29 (29) | 21 (23) | 27 (27) | 3 (3) | 8 (8) | 0 (0) | 0 (0)
Injection site cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 6 (6) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 6 (6) | 6 (6) | 11 (11) | 14 (15) | 15 (15) | 6 (6) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail bed infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 211 (238) | 251 (269) | 193 (209) | 208 (227) | 40 (43) | 36 (37) | 1 (1) | 1 (1)
Neuroborreliosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 6 (6) | 5 (5) | 7 (7) | 10 (10) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 35 (37) | 22 (23) | 25 (29) | 18 (18) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 3 (3) | 2 (3) | 10 (11) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Otitis externa fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 5 (5) | 5 (5) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parasitic gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perichondritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 22 (22) | 18 (18) | 30 (30) | 31 (34) | 5 (6) | 2 (2) | 1 (1) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 4 (4) | 9 (10) | 10 (10) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 17 (17) | 7 (7) | 17 (17) | 9 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 17 (20) | 22 (24) | 19 (19) | 18 (19) | 6 (6) | 4 (4) | 0 (0) | 0 (0)
Rhinolaryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 24 (25) | 26 (26) | 30 (31) | 22 (23) | 5 (5) | 9 (9) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tinea manuum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 5 (5) | 4 (4) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 7 (7) | 8 (8) | 5 (5) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 6 (6) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Toxoplasmosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 100 (107) | 75 (79) | 89 (96) | 77 (85) | 24 (24) | 14 (15) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 27 (27) | 36 (37) | 39 (41) | 40 (41) | 18 (18) | 11 (12) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 6 (6) | 8 (8) | 10 (10) | 6 (6) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aqueous humour leakage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 8 (8) | 6 (6) | 14 (14) | 8 (8) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 8 (8) | 13 (13) | 12 (13) | 8 (8) | 4 (4) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crush injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 3 (5) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 8 (8) | 9 (9) | 5 (5) | 5 (5) | 4 (5) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 5 (5) | 4 (4) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 8 (8) | 12 (12) | 7 (7) | 9 (9) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 8 (8) | 7 (7) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 6 (6) | 3 (3) | 8 (8) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Open fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic arthropathy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 7 (8) | 2 (2) | 7 (7) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood testosterone decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature fluctuation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 54 (57) | 2 (2) | 46 (53) | 2 (2) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Grip strength decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Precancerous cells present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 0 (0) | 16 (16) | 3 (3) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 5 (5) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 7 (7) | 3 (3) | 11 (11) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeding disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 13 (15) | 4 (4) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 7 (7) | 10 (10) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 6 (6) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 8 (8) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 110 (120) | 68 (73) | 99 (107) | 73 (86) | 22 (22) | 18 (20) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 4 (5) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 89 (95) | 63 (69) | 76 (85) | 82 (90) | 26 (27) | 27 (32) | 0 (0) | 1 (1)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 7 (7) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (5) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iliolumbar syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (10) | 8 (8) | 20 (22) | 12 (13) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (5) | 4 (4) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3) | 4 (5) | 4 (4) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 5 (6) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 40 (43) | 24 (26) | 44 (45) | 28 (28) | 3 (3) | 9 (9) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 13 (14) | 7 (7) | 6 (7) | 7 (7) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 243 (297) | 36 (43) | 177 (202) | 51 (56) | 32 (39) | 9 (11) | 2 (2) | 0 (0)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 32 (36) | 14 (15) | 24 (29) | 23 (25) | 4 (4) | 5 (5) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 19 (19) | 42 (44) | 44 (44) | 12 (13) | 6 (6) | 0 (0) | 2 (2)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 52 (55) | 44 (48) | 67 (80) | 40 (43) | 27 (29) | 14 (16) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (4) | 4 (5) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 4 (4) | 7 (7) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 4 (4) | 6 (7) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Benign ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 6 (6) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 4 (4) | 3 (3) | 6 (6) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 2 (2) | 2 (3) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 6 (6) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsions local (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 70 (78) | 34 (35) | 78 (80) | 60 (64) | 24 (25) | 15 (15) | 1 (1) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 5 (5) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial spasm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 5 (6) | 2 (2) | 5 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 475 (669) | 205 (275) | 329 (403) | 160 (212) | 61 (70) | 30 (36) | 1 (1) | 1 (2)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 6 (6) | 9 (11) | 12 (12) | 7 (7) | 3 (3) | 3 (3) | 1 (3) | 0 (0)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 9 (10) | 4 (4) | 12 (12) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 8 (15) | 3 (3) | 6 (6) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 13 (13) | 5 (5) | 9 (9) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 6 (6) | 6 (7) | 11 (11) | 20 (20) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Senile dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 13 (17) | 2 (2) | 17 (20) | 5 (6) | 5 (5) | 3 (4) | 0 (0) | 0 (0)
Spinal claudication (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stupor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 2 (2) | 5 (5) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 4 (4) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agoraphobia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 13 (13) | 3 (3) | 8 (8) | 11 (11) | 4 (4) | 6 (6) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aversion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 7 (7) | 9 (9) | 10 (11) | 4 (4) | 6 (6) | 0 (0) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphemia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphoria (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysthymic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Emotional disorder (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 34 (36) | 19 (23) | 29 (31) | 14 (14) | 9 (9) | 3 (3) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Listless (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obsessive thoughts (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychosomatic disease (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia, paranoid type (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis interstitial (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 5 (5) | 0 (0) | 4 (4) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 5 (5) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 8 (8) | 7 (7) | 8 (8) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital tract inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital ulceration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Male sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organic erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate induration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic disorder (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatism (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testis discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal erosion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 2 (2) | 9 (9) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 6 (6) | 5 (5) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 70 (74) | 64 (66) | 88 (92) | 96 (103) | 18 (18) | 22 (23) | 0 (0) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 8 (8) | 11 (11) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (6) | 5 (5) | 6 (7) | 1 (2) | 7 (12) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 12 (16) | 11 (11) | 7 (8) | 3 (3) | 2 (3) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 81 (84) | 64 (69) | 55 (56) | 56 (59) | 4 (4) | 12 (12) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural adhesion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 4 (5) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 4 (4) | 9 (9) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 11 (13) | 17 (19) | 14 (14) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 6 (6) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (3) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 4 (4) | 13 (13) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (4) | 5 (6) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (3) | 6 (6) | 7 (8) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 13 (13) | 23 (24) | 25 (26) | 24 (25) | 8 (8) | 7 (7) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 21 (22) | 7 (7) | 20 (20) | 14 (15) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 16 (16) | 4 (4) | 10 (10) | 8 (8) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 37 (38) | 35 (36) | 45 (48) | 56 (64) | 23 (24) | 13 (13) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (8) | 4 (4) | 9 (9) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 45 (46) | 40 (43) | 42 (44) | 63 (74) | 18 (20) | 9 (10) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 2 (2) | 9 (10) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Senile pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin warm (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 11 (11) | 6 (6) | 9 (9) | 13 (14) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occupational physical problem (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental implantation (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth cyst excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angiopathy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Behcet's syndrome (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure fluctuation (Surgical and medical procedures) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure inadequately controlled (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Essential hypertension (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Surgical and medical procedures) | 7 (8) | 0 (0) | 8 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Surgical and medical procedures) | 2 (2) | 2 (2) | 4 (4) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Haemorrhage (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Surgical and medical procedures) | 5 (5) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperaemia (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Surgical and medical procedures) | 25 (26) | 30 (30) | 36 (37) | 41 (41) | 8 (8) | 18 (19) | 1 (1) | 1 (1)
Hypertensive crisis (Surgical and medical procedures) | 0 (0) | 4 (4) | 4 (4) | 6 (8) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Surgical and medical procedures) | 2 (2) | 1 (1) | 7 (7) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haematoma (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemia (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labile blood pressure (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Orthostatic hypotension (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Surgical and medical procedures) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Raynaud's phenomenon (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporal arteritis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT03563183/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT03563183/SAP_001.pdf